CLINICAL TRIAL: NCT04748445
Title: Acute Respiratory Illness Surveillance (ARIS) by Monitoring Voice and Illness Symptom Changes Using a Mobile Application in a Low-Interventional Decentralized Study.
Brief Title: Acute Respiratory Illness Surveillance (AcRIS) With Mobile Application in a Low-Interventional Decentralized Study.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001293
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: Covid-19; Covid 19; Coronavirus; SARS-CoV-2; Flu; Influenza; RSV; Respiratory syncytial virus; Respiratory illness; Acute respiratory illness; remote trial; voice; AcRIS
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — SARS-CoV-2/Influenza/RSV RT-PCR
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants
  Interventions: Diagnostic Test: SARS-CoV-2/Influenza/RSV RT-PCR

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2/Influenza/RSV RT-PCR — nasal swab

SUMMARY:
The purpose of the AcRIS study is to obtain data to characterize the relationship between symptoms and voice features for (reverse transcription polymerase chain reaction (RT-PCR) confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), influenza virus, or Respiratory Syncytial Virus (RSV) positive participants with acute viral respiratory illness. This data will be used as the basis to build voice and symptom algorithm(s) for detection and monitoring of these illnesses. This would benefit vaccine development across several key disease areas, including SARS-CoV-2, influenza virus and RSV.

The study also models concepts of more efficient "flexible" clinical trials involving not only voice capture, but also web-based participant recruitment, enhanced participant engagement, and remote sample collection that could make future clinical studies more efficient. The clinical data obtained in this observational study could provide the documentation of the technology's performance needed to enable its deployment in future interventional studies.

DETAILED DESCRIPTION:
Each subject will be required to stay in the study for 6 weeks. If the participant tests positive for any of the three viruses at swab #1 or swab #2, they will continue the study until the end of Week 8.

Participants will record acute respiratory illnesses symptoms and voice data daily for up to a maximum of 8 weeks in both the well state and, should they become ill, the sick state, utilizing the Electronic diary on their Mobile application. Once enrolled, the participant will start recording symptoms and voice in the Electronic diary, with daily time commitment to this portion of the study expected to be 2-4 minutes. Two nasal self-swab collection kits will be ordered for delivery to the participant once they are enrolled in the study. The participant will be asked to self-swab when the test kit arrives (swab #1). The kit, including the specimen, will be returned to the central lab for RT-PCR SARS-CoV2/Influenza/RSV RT-PCR testing. The participant is expected to complete 3 phonemes and 5 lines of reading each day, in addition to score the self-reported symptoms in the Electronic diary. If participants become sick (self-report) with new or increased symptoms of acute respiratory illness symptoms, they will be asked to self-swab (swab #2) and return the sample for central SARS-CoV-2/Influenza/RSV RT-PCR testing. If the participant does not develop any new or increased symptoms between swab #1 and end of Week 6, they will obtain a self-swab (swab #2) at Day 42.

If the participant tests positive for any of the three viruses at swab #1 or swab #2, they will continue the study until end of week 8. If they test negative for the three viruses at swab #1 and swab #2, they will exit the study at approximately the end of week 6 when the test results are returned. The results of the RT-PCR testing will be shared with participants.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Age and Sex:

1. Male or female participants ≥18 years of age (or the minimum state specific age of consent if >18), at Screening visit.

   Type of Participant and Disease Characteristics:
2. Participants who are willing and able to comply with daily symptom and voice assessments on the electronic diary application and other study procedures, including self-collection of nasal swabs.
3. Expected to be available for the duration of the study.

Informed Consent:

4. Capable of giving signed informed consent

-

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Participants who self-report any medical condition, recreational substance use, or medication use which would prevent them from completing study tasks or impair the providing of informed consent, or in the investigator's judgment, make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
2. Participants who have been vaccinated with COVID-19 vaccine or are planning to get vaccinated during study participation.

   Participants can continue to use all other prescription or non-prescription medications.

   Prior/Concurrent Clinical Study Experience:
3. Previous vaccination with any licensed or investigational RSV vaccine or are planning to get vaccinated during study participation.
4. Previous administration with an investigational drug within 30 days of enrollment (or as determined by the local requirement) or planning to participate in an interventional trial during study conduct.

   Diagnostic Assessments:
5. Screening diagnostic assessments are not required for eligibility purposes.

   Other Exclusions:
6. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator including vendors, and their respective family members.
7. Participants who use a mobile device that does not meet the minimum requirements of the Electronic diary.
8. Participants who have previously been enrolled in the study cannot be re-enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Planned enrollment of approximately 8700 participants 18 years of age or older in order to have a total of N of 100 participants with (1) confirmed negative SARS-CoV-2, RSV or Influenza RT-PCR (swab #1) and (2) confirmed positive SARS-CoV-2 RT-PCR, influenza virus or RSV (swab #2) symptomatic completers.
Sampling Method: Non-Probability Sample
Enrollment: 9151 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Chappie K, Kell S, Qi D, Selig J, Christakis Y, Moreno X, Severson J, Best A, Wacnik P, Santamaria M, Zhang Y, Fry BA, Mather RJ. Comparing Phoneme Speech Recordings and Acoustic App Data Capture Experience for Android and iOS Mobile Device Users in the Large Decentralized AcRIS Study. J Voice. 2025 Jun 23:S0892-1997(25)00201-2. doi: 10.1016/j.jvoice.2025.05.016. Online ahead of print. PMID 40555587
- [Derived] Santamaria M, Christakis Y, Demanuele C, Zhang Y, Tuttle PG, Mamashli F, Bai J, Landman R, Chappie K, Kell S, Samuelsson JG, Talbert K, Seoane L, Mark Roberts W, Kabagambe EK, Capelouto J, Wacnik P, Selig J, Adamowicz L, Khan S, Mather RJ. Longitudinal voice monitoring in a decentralized Bring Your Own Device trial for respiratory illness detection. NPJ Digit Med. 2025 Apr 11;8(1):202. doi: 10.1038/s41746-025-01584-4. PMID 40210993
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=X9001293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational study involving collection of voice and respiratory symptoms data in participants in both the well state and sick state.
Groups:
- All Participants: Eligible participants aged 18 years and older recorded acute respiratory illnesses symptoms and voice data daily for up to a maximum of 8 weeks in both the well state and sick state, utilizing the electronic diary on their mobile application. Additionally, participants who performed two nasal self-swabs and the participants who tested positive for any of the three viruses (severe acute respiratory syndrome cornonavirus-2 [SARS-CoV-2], influenza virus and respiratory syncytial virus) at swab1 or swab 2, continued the study until end of Week 8. The participants who tested negative for the three viruses at swab 1 and swab 2, exited the study at end of Week 6.
Period: Overall Study
Arm/Group | All Participants
Started | 9151
Completed | 8520
Not Completed | 631
Not completed — No longer met eligibility criteria | 12
Not completed — Other | 36
Not completed — Withdrawal by Subject | 553
Not completed — Lost to Follow-up | 30

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who signed the informed consent document and were enrolled in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 9151
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.03 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7235
  Male | 1916
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 793
  Not Hispanic or Latino | 7915
  Unknown or Not Reported | 443
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 116
  Asian | 89
  Native Hawaiian or Other Pacific Islander | 18
  Black or African American | 1127
  White | 7112
  More than one race | 452
  Unknown or Not Reported | 237

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Self-Reported Symptom Scores From Well-to-Sick State Through Day 56
Description: Symptoms (fever, cough, difficult breathing, fatigue, runny nose, stuffy/blocked nose, sore throat, loss of taste/smell, chills, muscle pain, diarrhea, vomiting, headache, nausea, rigors, wheezing) recorded at least once daily in e-diary for 8 weeks & rated 0:none to 4:severe for fever & 0:none to 7:severe for other symptoms. Total symptom score=sum of all symptom scores in a recording session & mean of daily total symptom score=average across available sessions for each day, range=0 to 109, higher value=more severe total symptoms. Baseline=average of values up to 7 days before 1st occurrence of new/increased symptoms. If no data in 7 days, average of endpoint values for closest 3 days prior to 7 days used as baseline. Linear mixed effect model used for analysis for change from baseline in each symptom versus day during well to sick period, with slope (without intercept) included as fixed effects and random effects. Fixed effect of slope, as population level estimate, was reported.
Time Frame: Baseline up to Day 56
Population: Participants who initially were SARS-CoV-2, Influenza and/or RSV negative (at Swab 1) and had no acute symptoms, and became SARS-CoV-2, Influenza virus or RSV positive (at Swab 2) and symptomatic during the study were included. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 126
Scores on a scale
  Chills | 0.065 (0.0110)
  Cough | 0.281 (0.0361)
  Diarrhea | 0.036 (0.0077)
  Difficulty breathing | 0.113 (0.0263)
  Fatigue | 0.259 (0.0319)
  Fever | 0.029 (0.0050)
  Headache | 0.194 (0.0281)
  Loss of taste or smell | 0.103 (0.0266)
  Muscle pain | 0.181 (0.0268)
  Nausea | 0.044 (0.0096)
  Rigors | 0.030 (0.0085)
  Runny nose | 0.159 (0.0216)
  Sore throat | 0.222 (0.0330)
  Stuffy/blocked nose | 0.337 (0.0443)
  Vomiting | 0.005 (0.0017)
  Wheezing: number analyzed (Participants) | 121
  Wheezing | 0.049 (0.0174)
  Mean of daily total symptom score | 2.644 (0.3279)
Statistical Analysis 1: Comparison: All Participants; Chills; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.065, 90% CI 2-sided [0.046 to 0.083]
Statistical Analysis 2: Comparison: All Participants; Cough; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.281, 90% CI 2-sided [0.221 to 0.341]
Statistical Analysis 3: Comparison: All Participants; Diarrhea; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.036, 90% CI 2-sided [0.023 to 0.048]
Statistical Analysis 4: Comparison: All Participants; Difficulty breathing; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.113, 90% CI 2-sided [0.069 to 0.156]
Statistical Analysis 5: Comparison: All Participants; Fatigue; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.259, 90% CI 2-sided [0.206 to 0.312]
Statistical Analysis 6: Comparison: All Participants; Fever; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.029, 90% CI 2-sided [0.020 to 0.037]
Statistical Analysis 7: Comparison: All Participants; Headache; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.194, 90% CI 2-sided [0.148 to 0.241]
Statistical Analysis 8: Comparison: All Participants; Loss of taste or smell; Test type: Other; p = 0.0002, Mixed Models Analysis; Slope = 0.103, 90% CI 2-sided [0.059 to 0.148]
Statistical Analysis 9: Comparison: All Participants; Muscle pain; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.181, 90% CI 2-sided [0.137 to 0.226]
Statistical Analysis 10: Comparison: All Participants; Nausea; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.044, 90% CI 2-sided [0.028 to 0.060]
Statistical Analysis 11: Comparison: All Participants; Rigors; Test type: Other; p = 0.0007, Mixed Models Analysis; Slope = 0.030, 90% CI 2-sided [0.016 to 0.044]
Statistical Analysis 12: Comparison: All Participants; Runny nose; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.159, 90% CI 2-sided [0.123 to 0.195]
Statistical Analysis 13: Comparison: All Participants; Sore throat; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.222, 90% CI 2-sided [0.168 to 0.277]
Statistical Analysis 14: Comparison: All Participants; Stuffy/blocked nose; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.337, 90% CI 2-sided [0.264 to 0.411]
Statistical Analysis 15: Comparison: All Participants; Vomiting; Test type: Other; p = 0.0053, Mixed Models Analysis; Slope = 0.005, 90% CI 2-sided [0.002 to 0.007]
Statistical Analysis 16: Comparison: All Participants; Wheezing; Test type: Other; p = 0.0057, Mixed Models Analysis; Slope = 0.049, 90% CI 2-sided [0.020 to 0.078]
Statistical Analysis 17: Comparison: All Participants; Mean of daily total symptom score; Test type: Other; p < .0001, Mixed Models Analysis; Slope = 2.644, 90% CI 2-sided [2.101 to 3.188]

2. Primary Outcome: Change From Baseline in Voice Features (AHH_Max Phonation Time, EE_Jitter Local Absolute, MM_Jitter Local Absolute) Values From Well-to-Sick State Through Day 56
Description: Participants recorded voice features such as pitch, jitter once daily in an electronic diary for 8 weeks. Voice assessments were done by 2 phonemes: 'eee' and 'mmm' for 4 seconds (minimum 3 seconds), 1 phoneme: "ahh" sustained (as long as possible) and a 5-sentence reading passage. Max Phonation Time: duration that sound is held for. Jitter Local Absolute: average absolute difference between consecutive periods. Indicates how unsteady the pitch is across neighboring glottal pulses. Linear mixed effect model was used for analysis for change from baseline in each voice feature versus day during the well to sick period, with slope (without intercept) included as fixed effects and random effects. The fixed effect of the slope, as the population level estimate, was reported. The data given has exponential factor in addition to values mentioned. Individual exponential factors have been mentioned in respective row title.
Time Frame: Baseline up to Day 56
Population: Participants who initially were SARS-CoV-2, Influenza and/or RSV negative (at Swab 1) and had no acute symptoms, and became SARS-CoV-2, Influenza virus or RSV positive (at Swab 2) and symptomatic during the study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | All Participants
Number analyzed (Participants) | 126
Seconds
  AHH_Max Phonation Time: LSM (10^-1), SE (10^-2): number analyzed (Participants) | 124
  AHH_Max Phonation Time: LSM (10^-1), SE (10^-2) | -1.519 (2.769)
  EE_Jitter Local Absolute: LSM (10^-8) | 6.899 (0)
  MM_Jitter Local Absolute: LSM (10^-7) | -1.743 (0)
Statistical Analysis 1: Comparison: All Participants; AHH_Max Phonation Time (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and estimated value it was 10^-1. For dispersion value it was 10^-2); Test type: Other; p < .0001, Mixed Models Analysis; Slope = -1.519, 90% CI 2-sided [-1.978 to -1.060], Standard Error of Mean 2.769
Statistical Analysis 2: Comparison: All Participants; EE_Jitter Local Absolute (The statistical data given below have exponential factor in addition to the values mentioned. For estimated value it was 10^-8); Test type: Other; p < .0001, Mixed Models Analysis; Slope = 6.899, Standard Error of Mean 0
Statistical Analysis 3: Comparison: All Participants; MM_Jitter Local Absolute (The statistical data given below have exponential factor in addition to the values mentioned. For estimated value it was 10^-7); Test type: Other; p < .0001, Mixed Models Analysis; Slope = -1.743, Standard Error of Mean 0

3. Primary Outcome: Change From Baseline in Voice Feature (Cepstral Peak Prominence, Harmonicity, MFCC Mean, MFCC Std, SNR, Shimmer Local dB, Spectral Flatness, Third Octave Band, and VLHR) Values From Well-to-Sick State Through Day 56
Description: Harmonicity, flatness, shimmer recorded and assessed by phonemes: 'eee' and 'mmm' for 4 seconds, "ahh" sustained and 5-sentence reading passage. Cepstral Peak Prominence: voice quality measure. Harmonicity: degree of periodicity in signal. mel frequency cepstral coefficients (MFCC) mean: quantifies shape of spectrum. MFCC std: quantifies variation in spectral shape over time. Signal-to-noise ratio (SNR): how loud signal is compared to background. Shimmer Local dB: average absolute difference between amplitudes of consecutive periods (how unsteady sound intensity is across neighboring glottal pulses). Spectral Flatness: quantifies how tone-like a signal is based on spectral distribution. Third Octave Band: energy in 200 Hz third octave band relative to total. VLHR: degree of nasality. Linear mixed effect model used for analysis. Fixed effect of slope, as population level estimate is reported. Individual exponential factors for data presented have been mentioned in respective row title.
Time Frame: Baseline up to Day 56
Population: Participants who initially were SARS-CoV-2, Influenza and/or RSV negative (at Swab 1) and had no acute symptoms, and became SARS-CoV-2, Influenza virus or RSV positive (at Swab 2) and symptomatic during the study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Decibel
Arm/Group | All Participants
Number analyzed (Participants) | 126
Decibel
  EE_Cepstral Peak Prominence LSM (10^-3), SE (10^-2) | -1.326 (1.174)
  EE_Harmonicity LSM (10^-3), SE (10^-2) | 7.667 (1.741)
  EE_MFCC mean 01 LSM (10^0), SE (10^-1) | 1.268 (2.820)
  EE_MFCC mean 02 LSM (10^-1), SE (10^-1) | -1.752 (2.127)
  EE_MFCC mean 03 LSM (10^-1), SE (10^-1) | 1.390 (1.262)
  EE_MFCC mean 04 LSM (10^-1), SE (10^-1) | -1.407 (1.194)
  EE_MFCC mean 05 LSM (10^-3), SE (10^-2) | -4.466 (8.869)
  EE_MFCC mean 06 LSM (10^-1), SE (10^-2) | -1.572 (9.127)
  EE_MFCC mean 07 LSM (10^-1), SE (10^-2) | 1.248 (7.598)
  EE_MFCC mean 08 LSM (10^-1), SE (10^-2) | -1.054 (7.218)
  EE_MFCC mean 09 LSM (10^-2), SE (10^-2) | 5.944 (6.536)
  EE_MFCC mean 10 LSM (10^-2), SE (10^-2) | -3.115 (6.007)
  EE_MFCC mean 11 LSM (10^-2), SE (10^-2) | -1.908 (5.932)
  EE_MFCC mean 12 LSM (10^-4), SE (10^-2) | -6.574 (5.105)
  EE_MFCC mean 13 LSM (10^-3), SE (10^-2) | 5.026 (5.176)
  EE_MFCC std 01 LSM (10^-2), SE (10^-2) | 8.365 (2.873)
  EE_MFCC std 02 LSM (10^-2), SE (10^-2) | 2.906 (1.181)
  EE_MFCC std 03 LSM (10^-2), SE (10^-2) | 3.960 (1.447)
  EE_MFCC std 04 LSM (10^-2), SE (10^-2) | 2.816 (1.026)
  EE_MFCC std 05 LSM (10^-3), SE (10^-2) | 7.814 (1.034)
  EE_MFCC std 06 LSM (10^-2), SE (10^-3) | 1.151 (8.443)
  EE_MFCC std 07 LSM (10^-2), SE (10^-3) | 2.528 (8.228)
  EE_MFCC std 08 LSM (10^-2), SE (10^-3) | 1.755 (7.204)
  EE_MFCC std 09 LSM (10^-2), SE (10^-3) | 2.673 (5.892)
  EE_MFCC std 10 LSM (10^-2), SE (10^-3) | 1.394 (5.642)
  EE_MFCC std 11 LSM (10^-2), SE (10^-3) | 1.547 (6.666)
  EE_MFCC std 12 LSM (10^-2), SE (10^-3) | 1.118 (6.122)
  EE_MFCC std 13 LSM (10^-2), SE (10^-3) | 1.160 (5.226)
  EE_SNR LSM (10^-2), SE (10^-2) | 4.771 (3.351)
  EE_Shimmer Local dB LSM (10^-4), SE (10^-4) | 8.053 (9.807)
  EE_Spectral Flatness LSM (10^-2), SE (10^-2) | -3.945 (1.892)
  EE_Third Octave Band LSM (10^-2), SE (10^-2) | -7.075 (8.409)
  EE_VLHR LSM (10^-2), SE (10^-2) | 1.658 (3.607)
  MM_Cepstral Peak Prominence LSM (10^-2), SE (10^-2) | 1.172 (1.423)
  MM_Harmonicity LSM (10^-3), SE (10^-2) | -1.285 (2.112)
  MM_MFCC mean 01 LSM (10^-1), SE (10^-1) | 9.159 (2.641)
  MM_MFCC mean 02 LSM (10^-1), SE (10^-1) | -2.180 (1.894)
  MM_MFCC mean 03 LSM (10^-1), SE (10^-1) | 1.821 (1.028)
  MM_MFCC mean 04 LSM (10^-1), SE (10^-2) | -2.064 (8.474)
  MM_MFCC mean 05 LSM (10^-1), SE (10^-2) | -1.265 (9.670)
  MM_MFCC mean 06 LSM (10^-2), SE (10^-2) | 2.851 (9.960)
  MM_MFCC mean 07 LSM (10^-1), SE (10^-2) | 1.209 (7.569)
  MM_MFCC mean 08 LSM (10^-1), SE (10^-2) | -2.215 (8.498)
  MM_MFCC mean 09 LSM (10^-2), SE (10^-2) | 5.560 (7.072)
  MM_MFCC mean 10 LSM (10^-2), SE (10^-2) | 1.214 (6.190)
  MM_MFCC mean 11 LSM (10^-1), SE (10^-2) | -1.106 (4.852)
  MM_MFCC mean 12 LSM (10^-2), SE (10^-2) | -4.884 (4.827)
  MM_MFCC mean 13 LSM (10^-2), SE (10^-2) | 3.600 (5.634)
  MM_MFCC std 01 LSM (10^-2), SE (10^-2) | 2.909 (3.096)
  MM_MFCC std 02 LSM (10^-2), SE (10^-2) | 1.720 (2.595)
  MM_MFCC std 03 LSM (10^-3), SE (10^-2) | 4.403 (1.503)
  MM_MFCC std 04 LSM (10^-3), SE (10^-2) | 7.542 (1.639)
  MM_MFCC std 05 LSM (10^-2), SE (10^-3) | 2.386 (8.233)
  MM_MFCC std 06 LSM (10^-2), SE (10^-2) | 1.593 (1.243)
  MM_MFCC std 07 LSM (10^-3), SE (10^-2) | 2.902 (1.082)
  MM_MFCC std 08 LSM (10^-2), SE (10^-2) | 1.615 (1.118)
  MM_MFCC std 09 LSM (10^-2), SE (10^-2) | 1.116 (1.104)
  MM_MFCC std 10 LSM (10^-3), SE (10^-3) | -2.168 (9.632)
  MM_MFCC std 11 LSM (10^-2), SE (10^-2) | 1.394 (1.081)
  MM_MFCC std 12 LSM (10^-2), SE (10^-3) | 1.375 (6.622)
  MM_MFCC std 13 LSM (10^-3), SE (10^-2) | -2.892 (1.205)
  MM_SNR LSM (10^-3), SE (10^-2) | -3.105 (3.256)
  MM_Shimmer Local dB LSM (10^-4), SE (10^-4) | 6.145 (9.704)
  MM_Spectral Flatness LSM (10^-2), SE (10^-2) | -2.911 (1.969)
  MM_Third Octave Band LSM (10^-1), SE (10^-2) | -1.487 (8.770)
  MM_VLHR LSM (10^-3), SE (10^-2) | 3.089 (3.396)
  READ_MFCC mean 01 LSM (10^-1), SE (10^-1) | 8.362 (2.077)
  READ_MFCC mean 02 LSM (10^-2), SE (10^-1) | 3.559 (1.147)
  READ_MFCC mean 03 LSM (10^-1), SE (10^-2) | 2.043 (7.752)
  READ_MFCC mean 04 LSM (10^-2), SE (10^-2) | -8.280 (6.413)
  READ_MFCC mean 05 LSM (10^-2), SE (10^-2) | -2.415 (5.260)
  READ_MFCC mean 06 LSM (10^-1), SE (10^-2) | -1.209 (4.904)
  READ_MFCC mean 07 LSM (10^-2), SE (10^-2) | 2.617 (4.639)
  READ_MFCC mean 08 LSM (10^-2), SE (10^-2) | -7.305 (4.267)
  READ_MFCC mean 09 LSM (10^-2), SE (10^-2) | -2.369 (4.428)
  READ_MFCC mean 10 LSM (10^-2), SE (10^-2) | -7.377 (3.339)
  READ_MFCC mean 11 LSM (10^-3), SE (10^-2) | 8.703 (3.665)
  READ_MFCC mean 12 LSM (10^-2), SE (10^-2) | -7.414 (3.294)
  READ_MFCC mean 13 LSM (10^-2), SE (10^-2) | 2.929 (2.705)
  READ_MFCC std 01 LSM (10^-1), SE (10^-2) | -2.717 (6.612)
  READ_MFCC std 02 LSM (10^-2), SE (10^-2) | -5.798 (2.961)
  READ_MFCC std 03 LSM (10^-2), SE (10^-2) | -1.008 (1.778)
  READ_MFCC std 04 LSM (10^-2), SE (10^-2) | -2.230 (1.193)
  READ_MFCC std 05 LSM (10^-2), SE (10^-2) | -1.336 (1.176)
  READ_MFCC std 06 LSM (10^-3), SE (10^-2) | -6.497 (1.413)
  READ_MFCC std 07 LSM (10^-2), SE (10^-3) | -1.213 (7.700)
  READ_MFCC std 08 LSM (10^-3), SE (10^-3) | -7.959 (9.743)
  READ_MFCC std 09 LSM (10^-3), SE (10^-3) | -4.137 (8.017)
  READ_MFCC std 10 LSM (10^-4), SE (10^-3) | 3.760 (7.531)
  READ_MFCC std 11 LSM (10^-3), SE (10^-3) | -2.185 (5.703)
  READ_MFCC std 12 LSM (10^-3), SE (10^-3) | 7.716 (5.746)
  READ_MFCC std 13 LSM (10^-3), SE (10^-3) | -4.019 (6.419)
  READ_SNR LSM (10^-3), SE (10^-2) | 5.103 (2.737)
Statistical Analysis 1: Comparison: All Participants; EE_Cepstral Peak Prominence (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and dispersion value it was 10^-2. For estimated value it was 10^-3); Test type: Other; p = 0.9103, Mixed Models Analysis; Slope = -1.326, 90% CI 2-sided [-2.079 to 1.814], Standard Error of Mean 1.174
Statistical Analysis 2: Comparison: All Participants; EE_Harmonicity (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.6605, Mixed Models Analysis; Slope = 0.007667, 90% CI 2-sided [-0.02119 to 0.03653], Standard Error of Mean 1.741
Statistical Analysis 3: Comparison: All Participants; EE_MFCC mean 01 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-1); Test type: Other; p < .0001, Mixed Models Analysis; Slope = 1.268, 90% CI 2-sided [0.8012 to 1.736], Standard Error of Mean 2.820
Statistical Analysis 4: Comparison: All Participants; EE_MFCC mean 02 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-1); Test type: Other; p = 0.4117, Mixed Models Analysis; Slope = -1.752, 90% CI 2-sided [-5.276 to 1.773], Standard Error of Mean 2.127
Statistical Analysis 5: Comparison: All Participants; EE_MFCC mean 03 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-1. For lower limit it was 10^-2); Test type: Other; p = 0.2728, Mixed Models Analysis; Slope = 1.390, 90% CI 2-sided [-7.012 to 3.482], Standard Error of Mean 1.262
Statistical Analysis 6: Comparison: All Participants; EE_MFCC mean 04 (The statistical data given below have exponential factor in addition to the values mentioned. For lower limit, estimated value and dispersion value it was 10^-1. For upper limit it was 10^-2); Test type: Other; p = 0.2411, Mixed Models Analysis; Slope = -1.407, 90% CI 2-sided [-3.385 to 5.724], Standard Error of Mean 1.194
Statistical Analysis 7: Comparison: All Participants; EE_MFCC mean 05 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.9599, Mixed Models Analysis; Slope = -0.004466, 90% CI 2-sided [-0.1514 to 0.1425], Standard Error of Mean 8.869
Statistical Analysis 8: Comparison: All Participants; EE_MFCC mean 06 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0875, Mixed Models Analysis; Slope = -0.1572, 90% CI 2-sided [-0.3084 to -0.005942], Standard Error of Mean 9.127
Statistical Analysis 9: Comparison: All Participants; EE_MFCC mean 07 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit and estimated value it was 10^-1. For dispersion value it was 10^-2 and for lower limit it was 10^-3); Test type: Other; p = 0.1029, Mixed Models Analysis; Slope = 1.248, 90% CI 2-sided [-1.072 to 2.507], Standard Error of Mean 7.598
Statistical Analysis 10: Comparison: All Participants; EE_MFCC mean 08 (The statistical data given below have exponential factor in addition to the values mentioned. For lower limit and estimated value it was 10^-1. For upper limit and dispersion value it was 10^-2); Test type: Other; p = 0.1468, Mixed Models Analysis; Slope = -1.054, 90% CI 2-sided [-2.250 to 1.423], Standard Error of Mean 7.218
Statistical Analysis 11: Comparison: All Participants; EE_MFCC mean 09 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.3649, Mixed Models Analysis; Slope = 0.05944, 90% CI 2-sided [-0.04887 to 0.1678], Standard Error of Mean 6.536
Statistical Analysis 12: Comparison: All Participants; EE_MFCC mean 10 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.6050, Mixed Models Analysis; Slope = -0.03115, 90% CI 2-sided [-0.1307 to 0.06839], Standard Error of Mean 6.007
Statistical Analysis 13: Comparison: All Participants; EE_MFCC mean 11 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.7483, Mixed Models Analysis; Slope = -0.01908, 90% CI 2-sided [-0.1174 to 0.07922], Standard Error of Mean 5.932
Statistical Analysis 14: Comparison: All Participants; EE_MFCC mean 12 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and dispersion value it was 10^-2. For estimated value it was 10^-4); Test type: Other; p = 0.9897, Mixed Models Analysis; Slope = -6.574, 90% CI 2-sided [-8.526 to 8.394], Standard Error of Mean 5.105
Statistical Analysis 15: Comparison: All Participants; EE_MFCC mean 13 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and dispersion value it was 10^-2. For estimated value it was 10^-3); Test type: Other; p = 0.9228, Mixed Models Analysis; Slope = 5.026, 90% CI 2-sided [-8.074 to 9.080], Standard Error of Mean 5.176
Statistical Analysis 16: Comparison: All Participants; EE_MFCC std 01 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0043, Mixed Models Analysis; Slope = 0.08365, 90% CI 2-sided [0.03604 to 0.1313], Standard Error of Mean 2.873
Statistical Analysis 17: Comparison: All Participants; EE_MFCC std 02 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0153, Mixed Models Analysis; Slope = 0.02906, 90% CI 2-sided [0.009486 to 0.04863], Standard Error of Mean 1.181
Statistical Analysis 18: Comparison: All Participants; EE_MFCC std 03 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-2); Test type: Other; p = 0.0071, Mixed Models Analysis; Slope = 3.960, 90% CI 2-sided [1.563 to 6.357], Standard Error of Mean 1.447
Statistical Analysis 19: Comparison: All Participants; EE_MFCC std 04 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-2); Test type: Other; p = 0.0070, Mixed Models Analysis; Slope = 2.816, 90% CI 2-sided [1.115 to 4.516], Standard Error of Mean 1.026
Statistical Analysis 20: Comparison: All Participants; EE_MFCC std 05 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.4513, Mixed Models Analysis; Slope = 0.007814, 90% CI 2-sided [-0.009323 to 0.02495], Standard Error of Mean 1.034
Statistical Analysis 21: Comparison: All Participants; EE_MFCC std 06 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit and estimated value it was 10^-2. For lower limit and dispersion value it was 10^-3); Test type: Other; p = 0.1753, Mixed Models Analysis; Slope = 1.151, 90% CI 2-sided [-2.483 to 2.550], Standard Error of Mean 8.443
Statistical Analysis 22: Comparison: All Participants; EE_MFCC std 07 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and estimated value it was 10^-2. For dispersion it was 10^-3); Test type: Other; p = 0.0026, Mixed Models Analysis; Slope = 2.528, 90% CI 2-sided [1.164 to 3.891], Standard Error of Mean 8.228
Statistical Analysis 23: Comparison: All Participants; EE_MFCC std 08 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.0162, Mixed Models Analysis; Slope = 0.01755, 90% CI 2-sided [0.005616 to 0.02949], Standard Error of Mean 7.204
Statistical Analysis 24: Comparison: All Participants; EE_MFCC std 09 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and estimated value it was 10^-2. For dispersion value it was 10^-3); Test type: Other; p < .0001, Mixed Models Analysis; Slope = 2.673, 90% CI 2-sided [1.697 to 3.650], Standard Error of Mean 5.892
Statistical Analysis 25: Comparison: All Participants; EE_MFCC std 10 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.0148, Mixed Models Analysis; Slope = 0.01394, 90% CI 2-sided [0.004595 to 0.02329], Standard Error of Mean 5.642
Statistical Analysis 26: Comparison: All Participants; EE_MFCC std 11 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.0219, Mixed Models Analysis; Slope = 0.01547, 90% CI 2-sided [0.004425 to 0.02652], Standard Error of Mean 6.666
Statistical Analysis 27: Comparison: All Participants; EE_MFCC std 12 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit and estimated value it was 10^-2. For lower limit and dispersion value it was 10^-3); Test type: Other; p = 0.0703, Mixed Models Analysis; Slope = 1.118, 90% CI 2-sided [1.032 to 2.132], Standard Error of Mean 6.122
Statistical Analysis 28: Comparison: All Participants; EE_MFCC std 13 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.0282, Mixed Models Analysis; Slope = 0.01160, 90% CI 2-sided [0.002940 to 0.02026], Standard Error of Mean 5.226
Statistical Analysis 29: Comparison: All Participants; EE_SNR (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.1570, Mixed Models Analysis; Slope = 0.04771, 90% CI 2-sided [-0.007823 to 0.1032], Standard Error of Mean 3.351
Statistical Analysis 30: Comparison: All Participants; EE_Shimmer Local dB (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.4131, Mixed Models Analysis; Slope = 0.0008053, 90% CI 2-sided [-0.0008199 to 0.002431], Standard Error of Mean 9.807
Statistical Analysis 31: Comparison: All Participants; EE_Spectral Flatness (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0391, Mixed Models Analysis; Slope = -0.03945, 90% CI 2-sided [-0.07080 to -0.008096], Standard Error of Mean 1.892
Statistical Analysis 32: Comparison: All Participants; EE_Third Octave Band (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.4018, Mixed Models Analysis; Slope = -0.07075, 90% CI 2-sided [-0.2101 to 0.06860], Standard Error of Mean 8.409
Statistical Analysis 33: Comparison: All Participants; EE_VLHR (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-2); Test type: Other; p = 0.6466, Mixed Models Analysis; Slope = 1.658, 90% CI 2-sided [-4.319 to 7.635], Standard Error of Mean 3.607
Statistical Analysis 34: Comparison: All Participants; MM_Cepstral Peak Prominence (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-2); Test type: Other; p = 0.4118, Mixed Models Analysis; Slope = 1.172, 90% CI 2-sided [-1.186 to 3.530], Standard Error of Mean 1.423
Statistical Analysis 35: Comparison: All Participants; MM_Harmonicity (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and dispersion value it was 10^-2. For estimated value it was 10^-3); Test type: Other; p = 0.9481, Mixed Models Analysis; Slope = -1.282, 90% CI 2-sided [-3.385 to 3.129], Standard Error of Mean 1.965
Statistical Analysis 36: Comparison: All Participants; MM_MFCC mean 01 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-1); Test type: Other; p = 0.0007, Mixed Models Analysis; Slope = 0.9159, 90% CI 2-sided [0.4783 to 1.354], Standard Error of Mean 2.641
Statistical Analysis 37: Comparison: All Participants; MM_MFCC mean 02 (The statistical data given below have exponential factor in addition to the values mentioned. For lower limit, estimated value and dispersion value it was 10^-1. For upper limit it was 10^-2); Test type: Other; p = 0.2519, Mixed Models Analysis; Slope = -2.180, 90% CI 2-sided [-5.319 to 9.585], Standard Error of Mean 1.894
Statistical Analysis 38: Comparison: All Participants; MM_MFCC mean 03 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-1. For lower limit it was 10^-2); Test type: Other; p = 0.0791, Mixed Models Analysis; Slope = 1.821, 90% CI 2-sided [1.166 to 3.524], Standard Error of Mean 1.028
Statistical Analysis 39: Comparison: All Participants; MM_MFCC mean 04 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0163, Mixed Models Analysis; Slope = -0.2064, 90% CI 2-sided [-0.3468 to -0.06599], Standard Error of Mean 8.474
Statistical Analysis 40: Comparison: All Participants; MM_MFCC mean 05 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit and dispersion value it was 10^-2. For lower limit and estimated value it was 10^-1); Test type: Other; p = 0.1932, Mixed Models Analysis; Slope = -1.265, 90% CI 2-sided [-2.867 to 3.375], Standard Error of Mean 9.670
Statistical Analysis 41: Comparison: All Participants; MM_MFCC mean 06 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.7752, Mixed Models Analysis; Slope = 0.02851, 90% CI 2-sided [-0.1365 to 0.1936], Standard Error of Mean 9.960
Statistical Analysis 42: Comparison: All Participants; MM_MFCC mean 07 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit and estimated value it was 10^-1. For lower limit it was 10^-3. For dispersion value it was 10^-2); Test type: Other; p = 0.1126, Mixed Models Analysis; Slope = 1.209, 90% CI 2-sided [-4.480 to 2.464], Standard Error of Mean 7.569
Statistical Analysis 43: Comparison: All Participants; MM_MFCC mean 08 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0102, Mixed Models Analysis; Slope = -0.2215, 90% CI 2-sided [-0.3624 to -0.08072], Standard Error of Mean 8.498
Statistical Analysis 44: Comparison: All Participants; MM_MFCC mean 09 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.4332, Mixed Models Analysis; Slope = 0.05560, 90% CI 2-sided [-0.06159 to 0.1728], Standard Error of Mean 7.072
Statistical Analysis 45: Comparison: All Participants; MM_MFCC mean 10 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.8448, Mixed Models Analysis; Slope = 0.01214, 90% CI 2-sided [-0.09044 to 0.1147], Standard Error of Mean 6.190
Statistical Analysis 46: Comparison: All Participants; MM_MFCC mean 11 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0244, Mixed Models Analysis; Slope = -0.1106, 90% CI 2-sided [-0.1910 to -0.03016], Standard Error of Mean 4.852
Statistical Analysis 47: Comparison: All Participants; MM_MFCC mean 12 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.3136, Mixed Models Analysis; Slope = -0.04884, 90% CI 2-sided [-0.1288 to 0.03115], Standard Error of Mean 4.827
Statistical Analysis 48: Comparison: All Participants; MM_MFCC mean 13 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.5240, Mixed Models Analysis; Slope = 0.03600, 90% CI 2-sided [-0.05736 to 0.1294], Standard Error of Mean 5.634
Statistical Analysis 49: Comparison: All Participants; MM_MFCC std 01 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-2); Test type: Other; p = 0.3493, Mixed Models Analysis; Slope = 2.909, 90% CI 2-sided [-2.222 to 8.039], Standard Error of Mean 3.096
Statistical Analysis 50: Comparison: All Participants; MM_MFCC std 02 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-2); Test type: Other; p = 0.5087, Mixed Models Analysis; Slope = 1.720, 90% CI 2-sided [-2.580 to 6.019], Standard Error of Mean 2.595
Statistical Analysis 51: Comparison: All Participants; MM_MFCC std 03 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.7701, Mixed Models Analysis; Slope = 0.004403, 90% CI 2-sided [-0.02051 to 0.02931], Standard Error of Mean 1.503
Statistical Analysis 52: Comparison: All Participants; MM_MFCC std 04 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.6461, Mixed Models Analysis; Slope = 0.007542, 90% CI 2-sided [-0.01961 to 0.03470], Standard Error of Mean 1.639
Statistical Analysis 53: Comparison: All Participants; MM_MFCC std 05 (The statistical data given below have (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and estimated value it was 10^-2. For dispersion value it was 10^-3); Test type: Other; p = 0.0044, Mixed Models Analysis; Slope = 2.386, 90% CI 2-sided [1.022 to 3.750], Standard Error of Mean 8.233
Statistical Analysis 54: Comparison: All Participants; MM_MFCC std 06 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-2. For lower limit it was 10^-3); Test type: Other; p = 0.2022, Mixed Models Analysis; Slope = 1.593, 90% CI 2-sided [-4.663 to 3.652], Standard Error of Mean 1.243
Statistical Analysis 55: Comparison: All Participants; MM_MFCC std 07 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.7890, Mixed Models Analysis; Slope = 0.002902, 90% CI 2-sided [-0.01503 to 0.02084], Standard Error of Mean 1.082
Statistical Analysis 56: Comparison: All Participants; MM_MFCC std 08 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-2. For lower limit it was 10^-3); Test type: Other; p = 0.1510, Mixed Models Analysis; Slope = 1.615, 90% CI 2-sided [-2.371 to 3.467], Standard Error of Mean 1.118
Statistical Analysis 57: Comparison: All Participants; MM_MFCC std 09 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-2. For lower limit it was 10^-3); Test type: Other; p = 0.3138, Mixed Models Analysis; Slope = 1.116, 90% CI 2-sided [-7.126 to 2.945], Standard Error of Mean 1.104
Statistical Analysis 58: Comparison: All Participants; MM_MFCC std 10 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.8223, Mixed Models Analysis; Slope = -0.002168, 90% CI 2-sided [-0.01813 to 0.01379], Standard Error of Mean 9.632
Statistical Analysis 59: Comparison: All Participants; MM_MFCC std 11 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-2. For lower limit it was 10^-3); Test type: Other; p = 0.1997, Mixed Models Analysis; Slope = 1.394, 90% CI 2-sided [-3.978 to 3.185], Standard Error of Mean 1.081
Statistical Analysis 60: Comparison: All Participants; MM_MFCC std 12 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.0398, Mixed Models Analysis; Slope = 0.01375, 90% CI 2-sided [0.002780 to 0.02473], Standard Error of Mean 6.622
Statistical Analysis 61: Comparison: All Participants; MM_MFCC std 13 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.8107, Mixed Models Analysis; Slope = -0.002892, 90% CI 2-sided [-0.02286 to 0.01707], Standard Error of Mean 1.205
Statistical Analysis 62: Comparison: All Participants; MM_SNR (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and dispersion value it was 10^-2. For estimated value it was 10^-3); Test type: Other; p = 0.9242, Mixed Models Analysis; Slope = -3.105, 90% CI 2-sided [-5.706 to 5.085], Standard Error of Mean 3.256
Statistical Analysis 63: Comparison: All Participants; MM_Shimmer Local dB (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.5277, Mixed Models Analysis; Slope = 0.0006145, 90% CI 2-sided [-0.0009936 to 0.002223], Standard Error of Mean 9.704
Statistical Analysis 64: Comparison: All Participants; MM_Spectral Flatness (The statistical data given below have exponential factor in addition to the values mentioned. For lower limit, estimated value and dispersion value it was 10^-2. For upper limit it was 10^-3); Test type: Other; p = 0.1418, Mixed Models Analysis; Slope = -2.911, 90% CI 2-sided [-6.174 to 3.522], Standard Error of Mean 1.969
Statistical Analysis 65: Comparison: All Participants; MM_Third Octave Band (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0924, Mixed Models Analysis; Slope = -0.1487, 90% CI 2-sided [-0.2940 to -0.003375], Standard Error of Mean 8.770
Statistical Analysis 66: Comparison: All Participants; MM_VLHR (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and dispersion value it was 10^-2. For estimated value it was 10^-3); Test type: Other; p = 0.9277, Mixed Models Analysis; Slope = 3.089, 90% CI 2-sided [-5.318 to 5.936], Standard Error of Mean 3.396
Statistical Analysis 67: Comparison: All Participants; READ_MFCC mean 01 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-1); Test type: Other; p < .0001, Mixed Models Analysis; Slope = 0.8362, 90% CI 2-sided [0.4920 to 1.180], Standard Error of Mean 2.077
Statistical Analysis 68: Comparison: All Participants; READ_MFCC mean 02 (The statistical data given below have (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-1); Test type: Other; p = 0.7568, Mixed Models Analysis; Slope = 0.03559, 90% CI 2-sided [-0.1545 to 0.2256], Standard Error of Mean 1.147
Statistical Analysis 69: Comparison: All Participants; READ_MFCC mean 03 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0095, Mixed Models Analysis; Slope = 0.2043, 90% CI 2-sided [0.07585 to 0.3328], Standard Error of Mean 7.752
Statistical Analysis 70: Comparison: All Participants; READ_MFCC mean 04 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.1991, Mixed Models Analysis; Slope = -0.08280, 90% CI 2-sided [-0.1891 to 0.02348], Standard Error of Mean 6.413
Statistical Analysis 71: Comparison: All Participants; READ_MFCC mean 05 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.6469, Mixed Models Analysis; Slope = -0.02415, 90% CI 2-sided [-0.1113 to 0.06301], Standard Error of Mean 5.260
Statistical Analysis 72: Comparison: All Participants; READ_MFCC mean 06 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0150, Mixed Models Analysis; Slope = -0.1209, 90% CI 2-sided [-0.2022 to -0.03967], Standard Error of Mean 4.904
Statistical Analysis 73: Comparison: All Participants; READ_MFCC mean 07 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.5736, Mixed Models Analysis; Slope = 0.02617, 90% CI 2-sided [-0.05070 to 0.1030], Standard Error of Mean 4.639
Statistical Analysis 74: Comparison: All Participants; READ_MFCC mean 08 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0894, Mixed Models Analysis; Slope = -0.07305, 90% CI 2-sided [-0.1438 to -0.002335], Standard Error of Mean 4.267
Statistical Analysis 75: Comparison: All Participants; READ_MFCC mean 09 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-2); Test type: Other; p = 0.5936, Mixed Models Analysis; Slope = -2.369, 90% CI 2-sided [-9.706 to 4.968], Standard Error of Mean 4.428
Statistical Analysis 76: Comparison: All Participants; READ_MFCC mean 10 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0290, Mixed Models Analysis; Slope = -0.07377, 90% CI 2-sided [-0.1291 to -0.01844], Standard Error of Mean 3.339
Statistical Analysis 77: Comparison: All Participants; READ_MFCC mean 11 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.8127, Mixed Models Analysis; Slope = 0.008703, 90% CI 2-sided [-0.05203 to 0.06944], Standard Error of Mean 3.665
Statistical Analysis 78: Comparison: All Participants; READ_MFCC mean 12 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0262, Mixed Models Analysis; Slope = -0.07414, 90% CI 2-sided [-0.1287 to -0.01955], Standard Error of Mean 3.294
Statistical Analysis 79: Comparison: All Participants; READ_MFCC mean 13 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-2); Test type: Other; p = 0.2809, Mixed Models Analysis; Slope = 2.929, 90% CI 2-sided [-1.553 to 7.412], Standard Error of Mean 2.705
Statistical Analysis 80: Comparison: All Participants; READ_MFCC std 01 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and estimated value it was 10^-1. For dispersion value it was 10^-2); Test type: Other; p < .0001, Mixed Models Analysis; Slope = -2.717, 90% CI 2-sided [-3.812 to -1.621], Standard Error of Mean 6.612
Statistical Analysis 81: Comparison: All Participants; READ_MFCC std 02 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0524, Mixed Models Analysis; Slope = -0.05798, 90% CI 2-sided [-0.1070 to -0.008915], Standard Error of Mean 2.961
Statistical Analysis 82: Comparison: All Participants; READ_MFCC std 03 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-2); Test type: Other; p = 0.5716, Mixed Models Analysis; Slope = -1.008, 90% CI 2-sided [-3.955 to 1.938], Standard Error of Mean 1.778
Statistical Analysis 83: Comparison: All Participants; READ_MFCC std 04 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.0640, Mixed Models Analysis; Slope = -0.02230, 90% CI 2-sided [-0.04208 to -0.002526], Standard Error of Mean 1.193
Statistical Analysis 84: Comparison: All Participants; READ_MFCC std 05 (The statistical data given below have exponential factor in addition to the values mentioned. For lower limit, estimated value and dispersion value it was 10^-2. For upper limit it was 10^-3); Test type: Other; p = 0.2584, Mixed Models Analysis; Slope = -1.336, 90% CI 2-sided [-3.285 to 6.138], Standard Error of Mean 1.176
Statistical Analysis 85: Comparison: All Participants; READ_MFCC std 06 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.6465, Mixed Models Analysis; Slope = -0.006497, 90% CI 2-sided [-0.02992 to 0.01692], Standard Error of Mean 1.413
Statistical Analysis 86: Comparison: All Participants; READ_MFCC std 07 (The statistical data given below have exponential factor in addition to the values mentioned. For lower limit and estimated value it was 10^-2. For dispersion value it was 10^-3 and for upper limit it was 10^-4); Test type: Other; p = 0.1177, Mixed Models Analysis; Slope = -1.213, 90% CI 2-sided [-2.489 to 6.297], Standard Error of Mean 7.700
Statistical Analysis 87: Comparison: All Participants; READ_MFCC std 08 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.4155, Mixed Models Analysis; Slope = -0.007959, 90% CI 2-sided [-0.02411 to 0.008187], Standard Error of Mean 9.743
Statistical Analysis 88: Comparison: All Participants; READ_MFCC std 09 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.6067, Mixed Models Analysis; Slope = -0.004137, 90% CI 2-sided [-0.01742 to 0.009148], Standard Error of Mean 8.017
Statistical Analysis 89: Comparison: All Participants; READ_MFCC std 10 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.9603, Mixed Models Analysis; Slope = 0.0003760, 90% CI 2-sided [-0.01210 to 0.01286], Standard Error of Mean 7.531
Statistical Analysis 90: Comparison: All Participants; READ_MFCC std 11 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.7022, Mixed Models Analysis; Slope = -0.002185, 90% CI 2-sided [-0.01164 to 0.007265], Standard Error of Mean 5.703
Statistical Analysis 91: Comparison: All Participants; READ_MFCC std 12 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.1818, Mixed Models Analysis; Slope = 0.007716, 90% CI 2-sided [-0.001806 to 0.01724], Standard Error of Mean 5.746
Statistical Analysis 92: Comparison: All Participants; READ_MFCC std 13 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.5324, Mixed Models Analysis; Slope = -0.004019, 90% CI 2-sided [-0.01466 to 0.006618], Standard Error of Mean 6.419
Statistical Analysis 93: Comparison: All Participants; READ_SNR (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.8524, Mixed Models Analysis; Slope = 0.005103, 90% CI 2-sided [-0.04025 to 0.05046], Standard Error of Mean 2.737

4. Primary Outcome: Change From Baseline in Voice Feature (Coefficient of Variation, Mel Frequency Cepstral Coefficients (MFCC) 1st Order Delta, MFCC 2nd Order Delta) Values From Well-to-Sick State Through Day 56
Description: Voice features were recorded once daily in an electronic diary for 8 weeks. Assessments were done by 2 phonemes: 'eee' and 'mmm' for 4 seconds (minimum 3 seconds), 1 phoneme: "ahh" sustained (as long as possible) and a 5-sentence reading passage. Coefficient of Variation of F0: measures variation in pitch over time. MFCC 1st order delta: time-averaged estimate of first derivate of the MFCCs. MFCC 2nd order delta: time-averaged estimate of the second derivative of the MFCCs. Linear mixed effect model was used for analysis for change from baseline in each voice feature versus day during the well to sick period, with slope (without intercept) included as fixed effects and random effects. The fixed effect of the slope, as the population level estimate, was reported. The data given has exponential factor in addition to values mentioned. Individual exponential factors have been mentioned in respective row title.
Time Frame: Baseline up to Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Unitless
Arm/Group | All Participants
Number analyzed (Participants) | 126
Unitless
  EE_Coefficient of Variation F0 LSM (10^-4), SE (10^-4) | 2.975 (3.383)
  EE_MFCC 1st order delta 01 LSM (10^-3), SE (10^-3) | -5.601 (2.751)
  EE_MFCC 1st order delta 02 LSM (10^-3), SE (10^-3) | 4.120 (1.464)
  EE_MFCC 1st order delta 03 LSM (10^-3), SE (10^-3) | -3.067 (1.053)
  EE_MFCC 1st order delta 04 LSM (10^-3), SE (10^-4) | 2.780 (9.751)
  EE_MFCC 1st order delta 05 LSM (10^-3), SE (10^-4) | -1.324 (8.289)
  EE_MFCC 1st order delta 06 LSM (10^-4), SE (10^-4) | -2.606 (9.707)
  EE_MFCC 1st order delta 07 LSM (10^-4), SE (10^-4) | -5.071 (7.593)
  EE_MFCC 1st order delta 08 LSM (10^-4), SE (10^-4) | 3.067 (6.273)
  EE_MFCC 1st order delta 09 LSM (10^-3), SE (10^-4) | -1.649 (7.998)
  EE_MFCC 1st order delta 10 LSM (10^-4), SE (10^-4) | 8.236 (7.053)
  EE_MFCC 1st order delta 11 LSM (10^-4), SE (10^-4) | -2.920 (6.839)
  EE_MFCC 1st order delta 12 LSM (10^-4), SE (10^-4) | -3.363 (6.312)
  EE_MFCC 1st order delta 13 LSM (10^-4), SE (10^-4) | 7.281 (5.677)
  EE_MFCC 2nd order delta 01 LSM (10^-4), SE (10^-3) | 5.153 (1.523)
  EE_MFCC 2nd order delta 02 LSM (10^-3), SE (10^-4) | -1.330 (6.782)
  EE_MFCC 2nd order delta 03 LSM (10^-4), SE (10^-4) | -1.560 (6.763)
  EE_MFCC 2nd order delta 04 LSM (10^-5), SE (10^-4) | -9.713 (6.180)
  EE_MFCC 2nd order delta 05 LSM (10^-4), SE (10^-4) | 4.520 (5.576)
  EE_MFCC 2nd order delta 06 LSM (10^-4), SE (10^-4) | -1.528 (5.586)
  EE_MFCC 2nd order delta 07 LSM (10^-5), SE (10^-4) | -5.254 (4.217)
  EE_MFCC 2nd order delta 08 LSM (10^-4), SE (10^-4) | -4.591 (3.830)
  EE_MFCC 2nd order delta 09 LSM (10^-4), SE (10^-4) | 7.046 (3.687)
  EE_MFCC 2nd order delta 10 LSM (10^-4), SE (10^-4) | -1.564 (3.606)
  EE_MFCC 2nd order delta 11 LSM (10^-5), SE (10^-4) | 6.573 (2.810)
  EE_MFCC 2nd order delta 12 LSM (10^-4), SE (10^-4) | -4.071 (3.664)
  EE_MFCC 2nd order delta 13 LSM (10^-4), SE (10^-4) | 2.799 (3.317)
  MM_Coefficient of Variation F0 LSM (10^-4), SE (10^-4) | 1.123 (1.676)
  MM_MFCC 1st order delta 01 LSM (10^-5), SE (10^-3) | 7.586 (2.882)
  MM_MFCC 1st order delta 02 LSM (10^-4), SE (10^-3) | 8.249 (1.815)
  MM_MFCC 1st order delta 03 LSM (10^-3), SE (10^-3) | -1.188 (1.322)
  MM_MFCC 1st order delta 04 LSM (10^-4), SE (10^-3) | -7.258 (1.101)
  MM_MFCC 1st order delta 05 LSM (10^-3), SE (10^-4) | -1.326 (7.555)
  MM_MFCC 1st order delta 06 LSM (10^-4), SE (10^-3) | 5.502 (1.056)
  MM_MFCC 1st order delta 07 LSM (10^-4), SE (10^-4) | -4.691 (7.305)
  MM_MFCC 1st order delta 08 LSM (10^-3), SE (10^-4) | -1.530 (7.820)
  MM_MFCC 1st order delta 09 LSM (10^-4), SE (10^-4) | 4.166 (7.294)
  MM_MFCC 1st order delta 10 LSM (10^-3), SE (10^-4) | -2.112 (7.299)
  MM_MFCC 1st order delta 11 LSM (10^-4), SE (10^-4) | -7.706 (7.494)
  MM_MFCC 1st order delta 12 LSM (10^-4), SE (10^-4) | 2.388 (6.494)
  MM_MFCC 1st order delta 13 LSM (10^-4), SE (10^-4) | 2.121 (6.877)
  MM_MFCC 2nd order delta 01 LSM (10^-3), SE (10^-3) | -2.784 (1.667)
  MM_MFCC 2nd order delta 02 LSM (10^-4), SE (10^-4) | -1.368 (9.117)
  MM_MFCC 2nd order delta 03 LSM (10^-3), SE (10^-4) | -1.551 (6.294)
  MM_MFCC 2nd order delta 04 LSM (10^-3), SE (10^-4) | 1.840 (7.343)
  MM_MFCC 2nd order delta 05 LSM (10^-3), SE (10^-4) | 1.290 (5.029)
  MM_MFCC 2nd order delta 06 LSM (10^-4), SE (10^-4) | -1.473 (5.891)
  MM_MFCC 2nd order delta 07 LSM (10^-4), SE (10^-4) | -5.556 (4.647)
  MM_MFCC 2nd order delta 08 LSM (10^-3), SE (10^-4) | 1.128 (5.339)
  MM_MFCC 2nd order delta 09 LSM (10^-4), SE (10^-4) | -3.297 (5.134)
  MM_MFCC 2nd order delta 10 LSM (10^-4), SE (10^-4) | -2.104 (3.528)
  MM_MFCC 2nd order delta 11 LSM (10^-4), SE (10^-4) | 5.126 (4.289)
  MM_MFCC 2nd order delta 12 LSM (10^-4), SE (10^-4) | 2.703 (4.094)
  MM_MFCC 2nd order delta 13 LSM (10^-4), SE (10^-4) | -2.020 (5.334)
  READ_MFCC 1st order delta 01 LSM (10^-3), SE (10^-4) | -2.660 (9.220)
  READ_MFCC 1st order delta 02 LSM (10^-4), SE (10^-4) | 6.490 (4.448)
  READ_MFCC 1st order delta 03 LSM (10^-4), SE (10^-4) | 1.355 (3.323)
  READ_MFCC 1st order delta 04 LSM (10^-5), SE (10^-4) | 7.664 (2.574)
  READ_MFCC 1st order delta 05 LSM (10^-4), SE (10^-4) | -1.708 (2.028)
  READ_MFCC 1st order delta 06 LSM (10^-4), SE (10^-4) | 2.510 (1.904)
  READ_MFCC 1st order delta 07 LSM (10^-4), SE (10^-4) | 2.393 (1.627)
  READ_MFCC 1st order delta 08 LSM (10^-4), SE (10^-4) | 4.111 (1.553)
  READ_MFCC 1st order delta 09 LSM (10^-5), SE (10^-4) | -4.151 (1.134)
  READ_MFCC 1st order delta 10 LSM (10^-4), SE (10^-4) | 1.593 (1.291)
  READ_MFCC 1st order delta 11 LSM (10^-4), SE (10^-5) | 1.893 (9.442)
  READ_MFCC 1st order delta 12 LSM (10^-4), SE (10^-5) | 1.380 (6.614)
  READ_MFCC 1st order delta 13 LSM (10^-4), SE (10^-4) | 1.166 (1.040)
  READ_MFCC 2nd order delta 01 LSM (10^-3), SE (10^-4) | -1.190 (5.790)
  READ_MFCC 2nd order delta 02 LSM (10^-4), SE (10^-4) | -4.504 (3.040)
  READ_MFCC 2nd order delta 03 LSM (10^-4), SE (10^-4) | 2.968 (3.334)
  READ_MFCC 2nd order delta 04 LSM (10^-5), SE (10^-4) | -7.963 (2.101)
  READ_MFCC 2nd order delta 05 LSM (10^-4), SE (10^-4) | 5.075 (1.878)
  READ_MFCC 2nd order delta 06 LSM (10^-4), SE (10^-4) | -1.880 (1.174)
  READ_MFCC 2nd order delta 07 LSM (10^-4), SE (10^-4) | 1.667 (1.164)
  READ_MFCC 2nd order delta 08 LSM (10^-4), SE (10^-5) | 1.531 (9.552)
  READ_MFCC 2nd order delta 09 LSM (10^-4), SE (10^-4) | 1.989 (1.076)
  READ_MFCC 2nd order delta 10 LSM (10^-5), SE (10^-5) | 5.573 (9.318)
  READ_MFCC 2nd order delta 11 LSM (10^-5), SE (10^-5) | 1.774 (8.677)
  READ_MFCC 2nd order delta 12 LSM (10^-5), SE (10^-5) | 7.327 (6.630)
  READ_MFCC 2nd order delta 13 LSM (10^-4), SE (10^-5) | 1.534 (9.067)
Statistical Analysis 1: Comparison: All Participants; EE_Coefficient of Variation F0 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4; Test type: Other; p = 0.3809, Mixed Models Analysis; Slope = 2.975, 90% CI 2-sided [-2.631 to 8.580], Standard Error of Mean 3.383
Statistical Analysis 2: Comparison: All Participants; EE_MFCC 1st order delta 01 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3; Test type: Other; p = 0.0438, Mixed Models Analysis; Slope = -0.005601, 90% CI 2-sided [-0.01016 to -0.001043], Standard Error of Mean 2.751
Statistical Analysis 3: Comparison: All Participants; EE_MFCC 1st order delta 02 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-3; Test type: Other; p = 0.0057, Mixed Models Analysis; Slope = 4.120, 90% CI 2-sided [1.694 to 6.546], Standard Error of Mean 1.464
Statistical Analysis 4: Comparison: All Participants; EE_MFCC 1st order delta 03 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-3; Test type: Other; p = 0.0042, Mixed Models Analysis; Slope = -3.067, 90% CI 2-sided [-4.811 to -1.323], Standard Error of Mean 1.053
Statistical Analysis 5: Comparison: All Participants; EE_MFCC 1st order delta 04 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and estimated value it was 10^-3. For dispersion value it was 10^-4); Test type: Other; p = 0.0051, Mixed Models Analysis; Slope = 2.780, 90% CI 2-sided [1.164 to 4.396], Standard Error of Mean 9.751
Statistical Analysis 6: Comparison: All Participants; EE_MFCC 1st order delta 05 (The statistical data given below have exponential factor in addition to the values mentioned. For lower limit and estimated value it was 10^-3. For upper limit it was 10^-5 and for dispersion value it was 10^-4); Test type: Other; p = 0.1128, Mixed Models Analysis; Slope = -1.324, 90% CI 2-sided [-2.698 to 4.973], Standard Error of Mean 8.289
Statistical Analysis 7: Comparison: All Participants; EE_MFCC 1st order delta 06 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.7888, Mixed Models Analysis; Slope = -0.0002606, 90% CI 2-sided [-0.001869 to 0.001348], Standard Error of Mean 9.707
Statistical Analysis 8: Comparison: All Participants; EE_MFCC 1st order delta 07 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.5055, Mixed Models Analysis; Slope = -0.0005071, 90% CI 2-sided [-0.001765 to 0.0007512], Standard Error of Mean 7.593
Statistical Analysis 9: Comparison: All Participants; EE_MFCC 1st order delta 08 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.6257, Mixed Models Analysis; Slope = 0.0003067, 90% CI 2-sided [-0.0007328 to 0.001346], Standard Error of Mean 6.273
Statistical Analysis 10: Comparison: All Participants; EE_MFCC 1st order delta 09 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0413, Mixed Models Analysis; Slope = -0.001649, 90% CI 2-sided [-0.002974 to -0.0003238], Standard Error of Mean 7.998
Statistical Analysis 11: Comparison: All Participants; EE_MFCC 1st order delta 10 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.2451, Mixed Models Analysis; Slope = 0.0008236, 90% CI 2-sided [-0.0003452 to 0.001992], Standard Error of Mean 7.053
Statistical Analysis 12: Comparison: All Participants; EE_MFCC 1st order delta 11 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.6702, Mixed Models Analysis; Slope = -0.0002920, 90% CI 2-sided [-0.001425 to 0.0008413], Standard Error of Mean 6.839
Statistical Analysis 13: Comparison: All Participants; EE_MFCC 1st order delta 12 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.5951, Mixed Models Analysis; Slope = -0.0003363, 90% CI 2-sided [-0.001382 to 0.0007097], Standard Error of Mean 6.312
Statistical Analysis 14: Comparison: All Participants; EE_MFCC 1st order delta 13 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.2020, Mixed Models Analysis; Slope = 0.0007281, 90% CI 2-sided [-0.0002126 to 0.001669], Standard Error of Mean 5.677
Statistical Analysis 15: Comparison: All Participants; EE_MFCC 2nd order delta 01 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.7356, Mixed Models Analysis; Slope = 0.0005153, 90% CI 2-sided [-0.002008 to 0.003038], Standard Error of Mean 1.523
Statistical Analysis 16: Comparison: All Participants; EE_MFCC 2nd order delta 02 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0522, Mixed Models Analysis; Slope = -0.001330, 90% CI 2-sided [-0.002453 to -0.0002057], Standard Error of Mean 6.782
Statistical Analysis 17: Comparison: All Participants; EE_MFCC 2nd order delta 03 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.8180, Mixed Models Analysis; Slope = -0.0001560, 90% CI 2-sided [-0.001277 to 0.0009647], Standard Error of Mean 6.763
Statistical Analysis 18: Comparison: All Participants; EE_MFCC 2nd order delta 04 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4; Test type: Other; p = 0.8754, Mixed Models Analysis; Slope = -0.0000971, 90% CI 2-sided [-0.001121 to 0.0009270], Standard Error of Mean 6.180
Statistical Analysis 19: Comparison: All Participants; EE_MFCC 2nd order delta 05 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.4192, Mixed Models Analysis; Slope = 0.0004520, 90% CI 2-sided [-0.0004721 to 0.001376], Standard Error of Mean 5.576
Statistical Analysis 20: Comparison: All Participants; EE_MFCC 2nd order delta 06 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.7849, Mixed Models Analysis; Slope = -0.0001528, 90% CI 2-sided [-0.001079 to 0.0007729], Standard Error of Mean 5.586
Statistical Analysis 21: Comparison: All Participants; EE_MFCC 2nd order delta 07 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and dispersion value it was 10^-4. For estimated value it was 10^-5); Test type: Other; p = 0.9010, Mixed Models Analysis; Slope = -5.254, 90% CI 2-sided [-7.513 to 6.463], Standard Error of Mean 4.217
Statistical Analysis 22: Comparison: All Participants; EE_MFCC 2nd order delta 08 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.2329, Mixed Models Analysis; Slope = -0.0004591, 90% CI 2-sided [-0.001094 to 0.0001755], Standard Error of Mean 3.830
Statistical Analysis 23: Comparison: All Participants; EE_MFCC 2nd order delta 09 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0583, Mixed Models Analysis; Slope = 0.0007046, 90% CI 2-sided [0.00009366 to 0.001315], Standard Error of Mean 3.687
Statistical Analysis 24: Comparison: All Participants; EE_MFCC 2nd order delta 10 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.6654, Mixed Models Analysis; Slope = -1.564, 90% CI 2-sided [-7.540 to 4.413], Standard Error of Mean 3.606
Statistical Analysis 25: Comparison: All Participants; EE_MFCC 2nd order delta 11 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.8154, Mixed Models Analysis; Slope = 0.00006573, 90% CI 2-sided [-0.0003998 to 0.0005313], Standard Error of Mean 2.810
Statistical Analysis 26: Comparison: All Participants; EE_MFCC 2nd order delta 12 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.2687, Mixed Models Analysis; Slope = -0.0004071, 90% CI 2-sided [-0.001014 to 0.0002001], Standard Error of Mean 3.664
Statistical Analysis 27: Comparison: All Participants; EE_MFCC 2nd order delta 13 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.4005, Mixed Models Analysis; Slope = 2.799, 90% CI 2-sided [-2.698 to 8.296], Standard Error of Mean 3.317
Statistical Analysis 28: Comparison: All Participants; MM_Coefficient of Variation F0 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.5040, Mixed Models Analysis; Slope = 1.123, 90% CI 2-sided [-1.654 to 3.901], Standard Error of Mean 1.676
Statistical Analysis 29: Comparison: All Participants; MM_MFCC 1st order delta 01 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.9790, Mixed Models Analysis; Slope = 0.00007586, 90% CI 2-sided [-0.004701 to 0.004852], Standard Error of Mean 2.882
Statistical Analysis 30: Comparison: All Participants; MM_MFCC 1st order delta 02 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.6503, Mixed Models Analysis; Slope = 0.0008249, 90% CI 2-sided [-0.002183 to 0.003833], Standard Error of Mean 1.815
Statistical Analysis 31: Comparison: All Participants; MM_MFCC 1st order delta 03 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-3); Test type: Other; p = 0.3705, Mixed Models Analysis; Slope = -1.188, 90% CI 2-sided [-3.379 to 1.003], Standard Error of Mean 1.322
Statistical Analysis 32: Comparison: All Participants; MM_MFCC 1st order delta 04 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.5111, Mixed Models Analysis; Slope = -0.0007258, 90% CI 2-sided [-0.002551 to 0.001099], Standard Error of Mean 1.101
Statistical Analysis 33: Comparison: All Participants; MM_MFCC 1st order delta 05 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0816, Mixed Models Analysis; Slope = -0.001326, 90% CI 2-sided [-0.002578 to -0.0000744], Standard Error of Mean 7.555
Statistical Analysis 34: Comparison: All Participants; MM_MFCC 1st order delta 06 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.6034, Mixed Models Analysis; Slope = 0.0005502, 90% CI 2-sided [-0.001200 to 0.002301], Standard Error of Mean 1.056
Statistical Analysis 35: Comparison: All Participants; MM_MFCC 1st order delta 07 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.5220, Mixed Models Analysis; Slope = -0.0004691, 90% CI 2-sided [-0.001680 to 0.0007415], Standard Error of Mean 7.305
Statistical Analysis 36: Comparison: All Participants; MM_MFCC 1st order delta 08 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0526, Mixed Models Analysis; Slope = -0.001530, 90% CI 2-sided [-0.002826 to -0.0002344], Standard Error of Mean 7.820
Statistical Analysis 37: Comparison: All Participants; MM_MFCC 1st order delta 09 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.5689, Mixed Models Analysis; Slope = 0.0004166, 90% CI 2-sided [-0.0007920 to 0.001625], Standard Error of Mean 7.294
Statistical Analysis 38: Comparison: All Participants; MM_MFCC 1st order delta 10 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0045, Mixed Models Analysis; Slope = -0.002112, 90% CI 2-sided [-0.003321 to -0.0009020], Standard Error of Mean 7.299
Statistical Analysis 39: Comparison: All Participants; MM_MFCC 1st order delta 11 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.3058, Mixed Models Analysis; Slope = -0.0007706, 90% CI 2-sided [-0.002013 to 0.0004713], Standard Error of Mean 7.494
Statistical Analysis 40: Comparison: All Participants; MM_MFCC 1st order delta 12 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.7137, Mixed Models Analysis; Slope = 0.0002388, 90% CI 2-sided [-0.0008374 to 0.001315], Standard Error of Mean 6.494
Statistical Analysis 41: Comparison: All Participants; MM_MFCC 1st order delta 13 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.7583, Mixed Models Analysis; Slope = 0.0002121, 90% CI 2-sided [-0.0009275 to 0.001352], Standard Error of Mean 6.877
Statistical Analysis 42: Comparison: All Participants; MM_MFCC 2nd order delta 01 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit it was 10^-5. For lower limit, estimated value and dispersion value it was 10^-3); Test type: Other; p = 0.0974, Mixed Models Analysis; Slope = -2.784, 90% CI 2-sided [-5.547 to -2.155], Standard Error of Mean 1.667
Statistical Analysis 43: Comparison: All Participants; MM_MFCC 2nd order delta 02 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit and lower limit it was 10^-3. For estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.8810, Mixed Models Analysis; Slope = -1.368, 90% CI 2-sided [-1.648 to 1.374], Standard Error of Mean 9.117
Statistical Analysis 44: Comparison: All Participants; MM_MFCC 2nd order delta 03 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0151, Mixed Models Analysis; Slope = -0.001551, 90% CI 2-sided [-0.002594 to -0.0005077], Standard Error of Mean 6.294
Statistical Analysis 45: Comparison: All Participants; MM_MFCC 2nd order delta 04 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0135, Mixed Models Analysis; Slope = 0.001840, 90% CI 2-sided [0.0006233 to 0.003057], Standard Error of Mean 7.343
Statistical Analysis 46: Comparison: All Participants; MM_MFCC 2nd order delta 05 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0115, Mixed Models Analysis; Slope = 0.001290, 90% CI 2-sided [0.0004563 to 0.002123], Standard Error of Mean 5.029
Statistical Analysis 47: Comparison: All Participants; MM_MFCC 2nd order delta 06 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.8029, Mixed Models Analysis; Slope = -0.0001473, 90% CI 2-sided [-0.001123 to 0.0008288], Standard Error of Mean 5.891
Statistical Analysis 48: Comparison: All Participants; MM_MFCC 2nd order delta 07 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.2342, Mixed Models Analysis; Slope = -0.0005556, 90% CI 2-sided [-0.001326 to 0.0002146], Standard Error of Mean 4.647
Statistical Analysis 49: Comparison: All Participants; MM_MFCC 2nd order delta 08 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0366, Mixed Models Analysis; Slope = 0.001128, 90% CI 2-sided [0.0002436 to 0.002013], Standard Error of Mean 5.339
Statistical Analysis 50: Comparison: All Participants; MM_MFCC 2nd order delta 09 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.5220, Mixed Models Analysis; Slope = -0.0003297, 90% CI 2-sided [-0.001180 to 0.0005212], Standard Error of Mean 5.134
Statistical Analysis 51: Comparison: All Participants; MM_MFCC 2nd order delta 10 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.5520, Mixed Models Analysis; Slope = -2.104, 90% CI 2-sided [-7.950 to 3.742], Standard Error of Mean 3.528
Statistical Analysis 52: Comparison: All Participants; MM_MFCC 2nd order delta 11 (The statistical data given below have exponential factor in addition to the values mentioned. For ldispersion value it was 10^-4); Test type: Other; p = 0.2343, Mixed Models Analysis; Slope = 0.0005126, 90% CI 2-sided [-0.0001981 to 0.001223], Standard Error of Mean 4.289
Statistical Analysis 53: Comparison: All Participants; MM_MFCC 2nd order delta 12 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.5103, Mixed Models Analysis; Slope = 2.703, 90% CI 2-sided [-4.081 to 9.487], Standard Error of Mean 4.094
Statistical Analysis 54: Comparison: All Participants; MM_MFCC 2nd order delta 13 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.7056, Mixed Models Analysis; Slope = -0.0002020, 90% CI 2-sided [-0.001086 to 0.0006819], Standard Error of Mean 5.334
Statistical Analysis 55: Comparison: All Participants; READ_MFCC 1st order delta 01 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and dispersion value it was 10^-3. For estimated value it was 10^-4); Test type: Other; p = 0.0046, Mixed Models Analysis; Slope = -2.660, 90% CI 2-sided [-4.188 to -1.132], Standard Error of Mean 9.220
Statistical Analysis 56: Comparison: All Participants; READ_MFCC 1st order delta 02 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.1471, Mixed Models Analysis; Slope = 0.0006490, 90% CI 2-sided [-0.0000881 to 0.001386], Standard Error of Mean 4.448
Statistical Analysis 57: Comparison: All Participants; READ_MFCC 1st order delta 03 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.6842, Mixed Models Analysis; Slope = 1.355, 90% CI 2-sided [-4.152 to 6.862], Standard Error of Mean 3.323
Statistical Analysis 58: Comparison: All Participants; READ_MFCC 1st order delta 04 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.7664, Mixed Models Analysis; Slope = 0.00007664, 90% CI 2-sided [-0.0003499 to 0.0005032], Standard Error of Mean 2.574
Statistical Analysis 59: Comparison: All Participants; READ_MFCC 1st order delta 05 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.4015, Mixed Models Analysis; Slope = -1.708, 90% CI 2-sided [-5.069 to 1.654], Standard Error of Mean 2.028
Statistical Analysis 60: Comparison: All Participants; READ_MFCC 1st order delta 06 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-4. For lower limit it was 10^-5); Test type: Other; p = 0.1897, Mixed Models Analysis; Slope = 2.510, 90% CI 2-sided [-6.446 to 5.665], Standard Error of Mean 1.904
Statistical Analysis 61: Comparison: All Participants; READ_MFCC 1st order delta 07 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-4. For lower limit it was 10^-5); Test type: Other; p = 0.1439, Mixed Models Analysis; Slope = 2.393, 90% CI 2-sided [-3.035 to 5.090], Standard Error of Mean 1.627
Statistical Analysis 62: Comparison: All Participants; READ_MFCC 1st order delta 08 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.0092, Mixed Models Analysis; Slope = 4.111, 90% CI 2-sided [1.537 to 6.685], Standard Error of Mean 1.553
Statistical Analysis 63: Comparison: All Participants; READ_MFCC 1st order delta 09 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.7150, Mixed Models Analysis; Slope = -0.0000415, 90% CI 2-sided [-0.0002294 to 0.0001464], Standard Error of Mean 1.134
Statistical Analysis 64: Comparison: All Participants; READ_MFCC 1st order delta 10 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-4. For lower limit it was 10^-5); Test type: Other; p = 0.2194, Mixed Models Analysis; Slope = 1.593, 90% CI 2-sided [-5.457 to 3.731], Standard Error of Mean 1.291
Statistical Analysis 65: Comparison: All Participants; READ_MFCC 1st order delta 11 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-5); Test type: Other; p = 0.0471, Mixed Models Analysis; Slope = 0.0001893, 90% CI 2-sided [0.00003283 to 0.0003458], Standard Error of Mean 9.442
Statistical Analysis 66: Comparison: All Participants; READ_MFCC 1st order delta 12 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-5); Test type: Other; p = 0.0390, Mixed Models Analysis; Slope = 0.0001380, 90% CI 2-sided [0.00002840 to 0.0002476], Standard Error of Mean 6.614
Statistical Analysis 67: Comparison: All Participants; READ_MFCC 1st order delta 13 (The statistical data given below have (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-4. For lower limit it was 10^-5); Test type: Other; p = 0.2645, Mixed Models Analysis; Slope = 1.166, 90% CI 2-sided [-5.579 to 2.890], Standard Error of Mean 1.040
Statistical Analysis 68: Comparison: All Participants; READ_MFCC 2nd order delta 01 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0420, Mixed Models Analysis; Slope = -0.001190, 90% CI 2-sided [-0.002149 to -0.0002303], Standard Error of Mean 5.790
Statistical Analysis 69: Comparison: All Participants; READ_MFCC 2nd order delta 02 (The statistical data given below have exponential factor in addition to the values mentioned. For lower limit, estimated value and dispersion value it was 10^-4. For upper limit it was 10^-5); Test type: Other; p = 0.1410, Mixed Models Analysis; Slope = -4.504, 90% CI 2-sided [-9.542 to 5.341], Standard Error of Mean 3.040
Statistical Analysis 70: Comparison: All Participants; READ_MFCC 2nd order delta 03 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.3751, Mixed Models Analysis; Slope = 2.968, 90% CI 2-sided [-2.557 to 8.492], Standard Error of Mean 3.334
Statistical Analysis 71: Comparison: All Participants; READ_MFCC 2nd order delta 04 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.7053, Mixed Models Analysis; Slope = -0.0000796, 90% CI 2-sided [-0.0004277 to 0.0002685], Standard Error of Mean 2.101
Statistical Analysis 72: Comparison: All Participants; READ_MFCC 2nd order delta 05 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-4); Test type: Other; p = 0.0078, Mixed Models Analysis; Slope = 5.075, 90% CI 2-sided [1.964 to 8.187], Standard Error of Mean 1.878
Statistical Analysis 73: Comparison: All Participants; READ_MFCC 2nd order delta 06 (The statistical data given below have exponential factor in addition to the values mentioned. For lower limit, estimated value and dispersion value it was 10^-4. For upper limit it was 10^-6); Test type: Other; p = 0.1119, Mixed Models Analysis; Slope = -1.880, 90% CI 2-sided [-3.826 to 6.611], Standard Error of Mean 1.174
Statistical Analysis 74: Comparison: All Participants; READ_MFCC 2nd order delta 07 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^-4. For lower limit it was 10^-5); Test type: Other; p = 0.1545, Mixed Models Analysis; Slope = 1.667, 90% CI 2-sided [-2.615 to 3.596], Standard Error of Mean 1.164
Statistical Analysis 75: Comparison: All Participants; READ_MFCC 2nd order delta 08 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit and estimated value it was 10^-4. For lower limit it was 10^-6 and for dispersion value it was 10^-5); Test type: Other; p = 0.1114, Mixed Models Analysis; Slope = 1.531, 90% CI 2-sided [-5.164 to 3.114], Standard Error of Mean 9.552
Statistical Analysis 76: Comparison: All Participants; READ_MFCC 2nd order delta 09 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.0668, Mixed Models Analysis; Slope = 0.0001989, 90% CI 2-sided [0.00002067 to 0.0003772], Standard Error of Mean 1.076
Statistical Analysis 77: Comparison: All Participants; READ_MFCC 2nd order delta 10 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-5); Test type: Other; p = 0.5509, Mixed Models Analysis; Slope = 0.00005573, 90% CI 2-sided [-0.0000986 to 0.0002101], Standard Error of Mean 9.318
Statistical Analysis 78: Comparison: All Participants; READ_MFCC 2nd order delta 11 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-5); Test type: Other; p = 0.8383, Mixed Models Analysis; Slope = 0.00001774, 90% CI 2-sided [-0.0001260 to 0.0001615], Standard Error of Mean 8.677
Statistical Analysis 79: Comparison: All Participants; READ_MFCC 2nd order delta 12 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-5); Test type: Other; p = 0.2713, Mixed Models Analysis; Slope = 0.00007327, 90% CI 2-sided [-0.0000366 to 0.0001831], Standard Error of Mean 6.630
Statistical Analysis 80: Comparison: All Participants; READ_MFCC 2nd order delta 13 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-5); Test type: Other; p = 0.0931, Mixed Models Analysis; Slope = 0.0001534, 90% CI 2-sided [0.00000317 to 0.0003037], Standard Error of Mean 9.067

5. Primary Outcome: Change From Baseline in Voice Features (EE_Entropy, MM_Entropy) Values From Well-to-Sick State Through Day 56
Description: Participants recorded voice features such as entropy once daily in an electronic diary for 8 weeks. Voice assessments were done by 2 phonemes: 'eee' and 'mmm' for 4 seconds (minimum 3 seconds), 1 phoneme: "ahh" sustained (as long as possible) and a 5-sentence reading passage. Entropy: Shannon entropy of the spectral distribution. Quantifies tonailty similar to spectral flatness. "EE_Entropy" and "MM_Entropy" refer to this same measure computed on the "eee" and "mmm" phonemes, respectively. Linear mixed effect model was used for analysis for change from baseline in each voice feature versus day during the well to sick period, with slope (without intercept) included as fixed effects and random effects. The fixed effect of the slope, as the population level estimate, was reported. The data given has exponential factor in addition to values mentioned. Individual exponential factors have been mentioned in respective row title.
Time Frame: Baseline up to Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Bit
Arm/Group | All Participants
Number analyzed (Participants) | 126
Bit
  EE_Entropy: LSM (10^-3), SE (10^-3) | -1.931 (3.554)
  MM_Entropy: LSM (10^-4), SE (10^-3) | -1.479 (2.847)
Statistical Analysis 1: Comparison: All Participants; EE_Entropy (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, estimated value and dispersion value it was 10^-3); Test type: Other; p = 0.5878, Mixed Models Analysis; Slope = -1.931, 90% CI 2-sided [-7.820 to 3.958], Standard Error of Mean 3.554
Statistical Analysis 2: Comparison: All Participants; MM_Entropy (The statistical data given below have exponential factor in addition to the values mentioned. For estimated value it was 10^-4. For dispersion value, lower limit and upper limit it was 10^-3); Test type: Other; p = 0.9587, Mixed Models Analysis; Slope = -1.479, 90% CI 2-sided [-4.866 to 4.570], Standard Error of Mean 2.847

6. Primary Outcome: Change From Baseline in Voice Features (Formant and Formant Bandwidth) Values From Well-to-Sick State Through Day 56
Description: Participants recorded voice features once daily in an electronic diary for 8 weeks. Voice assessments were done by 2 phonemes: 'eee' and 'mmm' for 4 seconds (minimum 3 seconds), 1 phoneme: "ahh" sustained (as long as possible) and a 5-sentence reading passage. Formant: frequency at which the vocal tract produces an acoustic resonance. Formant Bandwidth: the spectral width of the acoustic resonance. Linear mixed effect model was used for analysis for change from baseline in each voice feature versus day during the well to sick period, with slope (without intercept) included as fixed effects and random effects. The fixed effect of the slope, as the population level estimate, was reported. The data given has exponential factor in addition to values mentioned. Individual exponential factors have been mentioned in respective row title.
Time Frame: Baseline up to Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Hertz
Arm/Group | All Participants
Number analyzed (Participants) | 126
Hertz
  EE_Formant 1: LSM (10^-2), SE (10^-1) | -3.262 (4.487)
  EE_Formant 1 Bandwidth: LSM (10^-2), SE (10^-1) | -6.912 (5.997)
  EE_Formant 2: LSM (10^-1), SE (10^0) | 1.985 (1.230)
  EE_Formant 2 Bandwidth: LSM (10^-1), SE (10^0) | 6.573 (2.191)
  EE_Formant 3: LSM (10^-1), SE (10^-1) | 6.504 (8.958)
  EE_Formant 3 Bandwidth: LSM (10^-2), SE (10^0) | 9.459 (1.255)
  MM_Formant 1: LSM (10^-1), SE (10^-1) | 6.945 (7.972)
  MM_Formant 1 Bandwidth: LSM (10^-2), SE (10^0) | 2.424 (1.021)
  MM_Formant 2: LSM (10^-1), SE (10^0) | -9.256 (1.083)
  MM_Formant 2 Bandwidth: LSM (10^-1), SE (10^0) | 9.350 (1.289)
  MM_Formant 3: LSM (10^0), SE (10^0) | 2.105 (1.231)
  MM_Formant 3 Bandwidth: LSM (10^0), SE (10^0) | 1.664 (1.358)
Statistical Analysis 1: Comparison: All Participants; EE_Formant 1 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and dispersion value it was 10^-1. For estimated value it was 10^-2); Test type: Other; p = 0.9421, Mixed Models Analysis; Slope = -3.262, 90% CI 2-sided [-7.761 to 7.109], Standard Error of Mean 4.487
Statistical Analysis 2: Comparison: All Participants; EE_Formant 1 Bandwidth (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-1); Test type: Other; p = 0.9084, Mixed Models Analysis; Slope = -0.06912, 90% CI 2-sided [-1.063 to 0.9247], Standard Error of Mean 5.997
Statistical Analysis 3: Comparison: All Participants; EE_Formant 2 (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit and dispersion value it was 10^0. For estimated value it was 10^-1); Test type: Other; p = 0.8721, Mixed Models Analysis; Slope = 1.985, 90% CI 2-sided [-1.841 to 2.238], Standard Error of Mean 1.230
Statistical Analysis 4: Comparison: All Participants; EE_Formant 2 Bandwidth (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^0); Test type: Other; p = 0.7647, Mixed Models Analysis; Slope = 0.6573, 90% CI 2-sided [-2.974 to 4.288], Standard Error of Mean 2.191
Statistical Analysis 5: Comparison: All Participants; EE_Formant 3 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-1); Test type: Other; p = 0.4692, Mixed Models Analysis; Slope = 0.6504, 90% CI 2-sided [-0.8341 to 2.135], Standard Error of Mean 8.958
Statistical Analysis 6: Comparison: All Participants; EE_Formant 3 Bandwidth (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^0); Test type: Other; p = 0.9400, Mixed Models Analysis; Slope = -0.09459, 90% CI 2-sided [-2.174 to 1.985], Standard Error of Mean 1.255
Statistical Analysis 7: Comparison: All Participants; MM_Formant 1 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-1); Test type: Other; p = 0.3853, Mixed Models Analysis; Slope = 0.6945, 90% CI 2-sided [-0.6265 to 2.015], Standard Error of Mean 7.972
Statistical Analysis 8: Comparison: All Participants; MM_Formant 1 Bandwidth (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^0); Test type: Other; p = 0.9811, Mixed Models Analysis; Slope = 0.02424, 90% CI 2-sided [-1.667 to 1.716], Standard Error of Mean 1.021
Statistical Analysis 9: Comparison: All Participants; MM_Formant 2 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^0); Test type: Other; p = 0.3944, Mixed Models Analysis; Slope = -0.9256, 90% CI 2-sided [-2.720 to 0.8690], Standard Error of Mean 1.083
Statistical Analysis 10: Comparison: All Participants; MM_Formant 2 Bandwidth (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^0); Test type: Other; p = 0.4696, Mixed Models Analysis; Slope = 0.9350, 90% CI 2-sided [-1.201 to 3.071], Standard Error of Mean 1.289
Statistical Analysis 11: Comparison: All Participants; MM_Formant 3 (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^0); Test type: Other; p = 0.0896, Mixed Models Analysis; Slope = 2.105, 90% CI 2-sided [0.06596 to 4.145], Standard Error of Mean 1.231
Statistical Analysis 12: Comparison: All Participants; MM_Formant 3 Bandwidth (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, estimated value and dispersion value it was 10^0. For lower limit it was 10^-1); Test type: Other; p = 0.2227, Mixed Models Analysis; Slope = 1.664, 90% CI 2-sided [-5.864 to 3.915], Standard Error of Mean 1.358

7. Primary Outcome: Change From Baseline in Voice Features (EE_Voiced Frames, MM_Voiced Frames) Values From Well-to-Sick State Through Day 56
Description: Participants recorded voice features once daily in an electronic diary for 8 weeks. Voice assessments were done by 2 phonemes: 'eee' and 'mmm' for 4 seconds (minimum 3 seconds), 1 phoneme: "ahh" sustained (as long as possible) and a 5-sentence reading passage. The voiced frames rate indicates how much of the sound is voiced. EE and MM refer to the sounds on which the measure is computed. Linear mixed effect model was used for analysis for change from baseline in each voice feature versus day during the well to sick period, with slope (without intercept) included as fixed effects and random effects. The fixed effect of the slope, as the population level estimate, was reported. The data given has exponential factor in addition to values mentioned. Individual exponential factors have been mentioned in respective row title.
Time Frame: Baseline up to Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Frame per second
Arm/Group | All Participants
Number analyzed (Participants) | 126
Frame per second
  EE_Voiced Frames: LSM (10^-4), SE (10^-3) | -4.024 (3.122)
  MM_Voiced Frames: LSM (10^-4), SE (10^-4) | -6.624 (7.961)
Statistical Analysis 1: Comparison: All Participants; EE_Voiced Frames (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, and dispersion value it was 10^-3. For estimated value it was 10^-4); Test type: Other; p = 0.8977, Mixed Models Analysis; Slope = -4.024, 90% CI 2-sided [-5.577 to 4.772], Standard Error of Mean 3.122
Statistical Analysis 2: Comparison: All Participants; MM_Voiced Frames (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-4); Test type: Other; p = 0.4070, Mixed Models Analysis; Slope = -0.0006624, 90% CI 2-sided [-0.001982 to 0.0006569], Standard Error of Mean 7.961

8. Primary Outcome: Change From Baseline in Voice Features (EE_Jitter Local, MM_Jitter Local) Values From Well-to-Sick State Through Day 56
Description: Voice features such as jitter were recorded once daily in an electronic diary for 8 weeks. Voice assessments were done by 2 phonemes: 'eee' and 'mmm' for 4 seconds (minimum 3 seconds), 1 phoneme: "ahh" sustained (as long as possible) and a 5-sentence reading passage. Jitter Local: average absolute difference between consecutive periods divided by the average period as a percentage. Indicates how unsteady the pitch is across neighboring glottal pulses. Linear mixed effect model was used for analysis for change from baseline in each voice feature versus day during the well to sick period, with slope (without intercept) included as fixed effects and random effects. The fixed effect of the slope, as the population level estimate, was reported. The data given has exponential factor in addition to values mentioned. Individual exponential factors have been mentioned in respective row title.
Time Frame: Baseline up to Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of period
Arm/Group | All Participants
Number analyzed (Participants) | 126
Percentage of period
  EE_Jitter Local: LSM (10^-4), SE (10^-3) | 8.654 (1.441)
  MM_Jitter Local: LSM (10^-4), SE (10^-3) | -2.206 (3.176)
Statistical Analysis 1: Comparison: All Participants; EE_Jitter Local (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-3); Test type: Other; p = 0.5491, Mixed Models Analysis; Slope = 0.0008654, 90% CI 2-sided [-0.001522 to 0.003253], Standard Error of Mean 1.441
Statistical Analysis 2: Comparison: All Participants; MM_Jitter Local (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, and dispersion value it was 10^-3. For estimated value it was 10^-4); Test type: Other; p = 0.9447, Mixed Models Analysis; Slope = -2.206, 90% CI 2-sided [-5.483 to 5.042], Standard Error of Mean 3.176

9. Primary Outcome: Change From Baseline in Voice Features (EE_Shimmer Local, MM_Shimmer Local) Values From Well-to-Sick State Through Day 56
Description: Voice features such as shimmer were once daily in an electronic diary for 8 weeks. Voice assessments were done by 2 phonemes: 'eee' and 'mmm' for 4 seconds (minimum 3 seconds), 1 phoneme: "ahh" sustained (as long as possible) and a 5-sentence reading passage. Shimmer Local: average absolute difference between the amplitudes of consecutive periods divided by the average amplitude as a percentage. Indicates how unsteady the sound intensity is across neighboring glottal pulses. Linear mixed effect model was used for analysis for change from baseline in each voice feature versus day during the well to sick period, with slope (without intercept) included as fixed effects and random effects. The fixed effect of the slope, as the population level estimate, was reported. The data given has exponential factor in addition to values mentioned. Individual exponential factors have been mentioned in respective row title.
Time Frame: Baseline up to Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of amplitude
Arm/Group | All Participants
Number analyzed (Participants) | 126
Percentage of amplitude
  EE_Shimmer Local: LSM (10^-3), SE (10^-2) | 7.567 (1.120)
  MM_Shimmer Local: LSM (10^-3), SE (10^-2) | 6.060 (1.101)
Statistical Analysis 1: Comparison: All Participants; EE_Shimmer Local (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.5004, Mixed Models Analysis; Slope = 0.007567, 90% CI 2-sided [-0.01099 to 0.02612], Standard Error of Mean 1.120
Statistical Analysis 2: Comparison: All Participants; MM_Shimmer Local (The statistical data given below have exponential factor in addition to the values mentioned. For dispersion value it was 10^-2); Test type: Other; p = 0.5831, Mixed Models Analysis; Slope = 0.006060, 90% CI 2-sided [-0.01219 to 0.02431], Standard Error of Mean 1.101

10. Primary Outcome: Change From Baseline in Voice Features (READ_Speaking Rate) Values From Well-to-Sick State Through Day 56
Description: Participants recorded voice features once daily in an electronic diary for 8 weeks. Voice assessments were done by 2 phonemes: 'eee' and 'mmm' for 4 seconds (minimum 3 seconds), 1 phoneme: "ahh" sustained (as long as possible) and a 5-sentence reading passage. Baseline was average of endpoint values up to 7 days before first occurrence of new/increased symptoms. If participant had no data in 7 days, average of endpoint values for closest 3 days prior to these 7 days was used as baseline. Linear mixed effect model was used for analysis for change from baseline in each voice feature versus day during the well to sick period, with slope (without intercept) included as fixed effects and random effects. The fixed effect of the slope, as the population level estimate, was reported. The data given has exponential factor (i.e. LSM*10^-2, SE*10^-3) in addition to values mentioned.
Time Frame: Baseline up to Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Syllable per second
Arm/Group | All Participants
Number analyzed (Participants) | 126
Syllable per second | 2.130 (3.211)
Statistical Analysis 1: Comparison: All Participants; READ_Speaking Rate (The statistical data given below have exponential factor in addition to the values mentioned. For upper limit, lower limit, and estimated value it was 10^-2. For dispersion value it was 10^-3); Test type: Other; p < .0001, Mixed Models Analysis; Slope = 2.130, 90% CI 2-sided [1.598 to 2.662], Standard Error of Mean 3.211

11. Secondary Outcome: Percentage of Compliant Days in Total Days of Symptoms and Total Days of Voice Recordings Entered in the Electronic Diary
Description: In this outcome measure, percentage of compliant days in total days of self-reported symptoms and total days of voice recordings as entered in the electronic diary were reported. Compliant days were calculated for the following and expressed as percentage: symptom compliance = number of compliant days of self-reported symptoms divided by the total number of days in the study. Voice compliance (expressed as percentage) = number of compliant days of completed voice recordings divided by the total number of days in the study. Partial voice compliance (expressed as percentage) = number of compliant days of partially completed voice recordings divided by the total number of days in the study. Symptom and voice compliance (expressed as percentage) = number of compliant days of self-reported symptoms and completed voice recordings divided by the total number of days in the study. Participants who experienced technical issues due to study operational errors were excluded.
Time Frame: Day 1 up to Day 56
Population: Full analysis set included all participants who signed the informed consent document and enrolled in the study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | All Participants
Number analyzed (Participants) | 8755
Percentage of days
  Symptom Compliance | 33.81 (35.158)
  Voice Compliance | 32.06 (34.535)
  Partial Voice Compliance | 0.49 (1.369)
  Symptom and Voice Compliance | 32.06 (34.535)

12. Secondary Outcome: Percentage of Quality Voice Recordings
Description: In this outcome measure, percentage was calculated over the number of days that the participant was able to complete the task for each recording. Participants were required to record their daily voice in electronic diary and the assessment included 2 phonemes: 'eee' and 'mmm' for 4 seconds (minimum 3 seconds), 1 phoneme: "ahh" sustained (as long as possible) and a 5-sentence reading passage. Quality recordings were defined as recordings exceeding signal-to-noise (SNR) and duration thresholds (i.e. SNR >= 20 decibels [dB] that have duration >= 3 seconds for phoneme and >= 10 seconds for reading tasks). In the case of multiple electronic diary sessions per day, the session with the highest quality voice recordings for that day was used in this analysis.
Time Frame: Day 1 up to Day 56
Population: Full analysis set included all participants who signed the informed consent document and enrolled in the study.
Measure: Mean (Standard Deviation); unit: Percentage of quality recordings
Arm/Group | All Participants
Number analyzed (Participants) | 9151
Percentage of quality recordings | 84.15 (20.23)

13. Secondary Outcome: Percentage of Participants With a Positive Self-Swab Result for SARS-CoV-2 and/or Influenza and/or RSV
Description: In this outcome measure, percentage of participants with valid self-swab 1 and 2 results positive for SARS-COV-2, Flu A, Flu B, RSV and SARS-CoV-2 and/or Influenza (Flu A/Flu B) and/or RSV were reported.
Time Frame: Day 2 up to Day 43
Population: Full analysis set included all participants who signed the informed consent document and enrolled in the study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 6259
Percentage of participants
  Self-swab 1: SARS-COV-2: number analyzed (Participants) | 3623
  Self-swab 1: SARS-COV-2 | 6
  Self-swab 1: Flu A: number analyzed (Participants) | 3623
  Self-swab 1: Flu A | 0.2
  Self-swab 1: Flu B: number analyzed (Participants) | 3623
  Self-swab 1: Flu B | 0
  Self-swab 1: RSV: number analyzed (Participants) | 3623
  Self-swab 1: RSV | 0.1
  Self-swab 1: SARS-CoV-2 and/or Influenza and/or RSV: number analyzed (Participants) | 3623
  Self-swab 1: SARS-CoV-2 and/or Influenza and/or RSV | 6.3
  Self-swab 2: SARS-COV-2: number analyzed (Participants) | 2636
  Self-swab 2: SARS-COV-2 | 7.7
  Self-swab 2: Flu A: number analyzed (Participants) | 2636
  Self-swab 2: Flu A | 0.2
  Self-swab 2: Flu B: number analyzed (Participants) | 2636
  Self-swab 2: Flu B | 0
  Self-swab 2: RSV: number analyzed (Participants) | 2636
  Self-swab 2: RSV | 0.6
  Self-swab 2: SARS-CoV-2 and/or Influenza and/or RSV: number analyzed (Participants) | 2636
  Self-swab 2: SARS-CoV-2 and/or Influenza and/or RSV | 8.5

14. Secondary Outcome: Percentage of Participants Who Administered Self-swab 1 and Self-swab 2
Description: In this outcome measure, percentage of participants who administered self-swab 1, self-swab 2 and self-swab 1 and 2 excluding participants who experienced technical issues due to study operational errors were reported.
Time Frame: Day 2 up to Day 43
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 8755
Percentage of participants
  Participants who administered self-swab 1 | 43.4
  Participants who administered self-swab 2 | 31.4
  Participants who administered self-swab 1 and self-swab 2 | 28.3

15. Secondary Outcome: Number of Days Between Reporting Symptoms and Recording Swab 2 in the Electronic-Diary
Description: In this outcome measure, number of days from symptom onset (reporting new or increased symptoms in the electronic diary) to the day of recording Swab 2 day in the electronic diary averaged across participants who administered self-swab 2 was reported.
Time Frame: Day 2 Up to Day 43
Population: Full analysis set included all participants who signed the informed consent document and enrolled in the study. Here, 'Overall Number of Participants Analyzed' signifies participants had administered self swab 2 and were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 1578
Days | 18.98 (17.01)

16. Secondary Outcome: Percentage of Participants Reporting Symptoms in the Electronic Diary Who Have a Self-swab Collected at or Around Symptom Onset
Description: In this outcome measure, 1) participants (par) who administered (adm) self-swab 2 (SS2) before Week 6 (W6) divided by the number of participants who reported new or increased (inc) symptoms (sym) in the electronic diary (e-diary) before W6 and 2) number of participants who reported new or increased symptoms in the e-diary before Week 6 divided by the number of participants who administered self-swab 2 before Week 6 were reported in percentage.
Time Frame: Day 2 Up to Day 43
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 2554
Percentage of participants
  Par who adm SS2 before W6/par who reported new or inc symptoms in e-diary before W6 | 9.3
  Par who reported new or inc sym in e-diary before W6/par who adm SS2 before W6: number analyzed (Participants) | 1065
  Par who reported new or inc sym in e-diary before W6/par who adm SS2 before W6 | 22.3

17. Secondary Outcome: Percentage of Participants Who Administered Self-swabs With Valid Results
Description: In this outcome measure, percentage of participants with valid (positive or negative) self-swab results for SARS-CoV-2, Flu A, Flu b and RSV were reported.
Time Frame: Day 2 Up to Day 43
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 6788
Percentage of participants
  Positive or negative self-swab 1 result for SARS-CoV-2: number analyzed (Participants) | 3971
  Positive or negative self-swab 1 result for SARS-CoV-2 | 91.24
  Positive or negative self-swab 1 result for Flu A: number analyzed (Participants) | 3971
  Positive or negative self-swab 1 result for Flu A | 91.21
  Positive or negative self-swab 1 result for Flu B: number analyzed (Participants) | 3971
  Positive or negative self-swab 1 result for Flu B | 91.21
  Positive or negative self-swab 1 result for RSV: number analyzed (Participants) | 3971
  Positive or negative self-swab 1 result for RSV | 91.21
  Positive or negative self-swab 2 result for SARS-CoV-2: number analyzed (Participants) | 2817
  Positive or negative self-swab 2 result for SARS-CoV-2 | 93.57
  Positive or negative self-swab 2 result for Flu A: number analyzed (Participants) | 2817
  Positive or negative self-swab 2 result for Flu A | 93.57
  Positive or negative self-swab 2 result for Flu B: number analyzed (Participants) | 2817
  Positive or negative self-swab 2 result for Flu B | 93.57
  Positive or negative self-swab 2 result for RSV: number analyzed (Participants) | 2817
  Positive or negative self-swab 2 result for RSV | 93.57

ADVERSE EVENTS:
Time Frame: Maximum up to Day 56
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/9151
Serious Adverse Events (participants affected / at risk) | 0/9151
Other Adverse Events (participants affected / at risk) | 28/9151
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=9151)
Lacrimation increased (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Chills (General disorders) | 4
Fatigue (General disorders) | 4
Malaise (General disorders) | 1
Pain (General disorders) | 5
Pyrexia (General disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 11
Migraine (Nervous system disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT04748445/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04748445/SAP_001.pdf